#### 1 TITLE PAGE



VERTEX PHARMACEUTICALS INCORPORATED

# Clinical Study Protocol

A Phase 3, Randomized, Double-blind, Controlled Study Evaluating the Efficacy and Safety of VX-659 Combination Therapy in Subjects With Cystic Fibrosis Who Are Homozygous for the *F508del* Mutation (F/F)

Vertex Study Number: VX17-659-103

EudraCT Number: 2017-004133-82

**Date of Protocol:** 27 April 2018 (Version 3.0)

Vertex Pharmaceuticals Incorporated 50 Northern Avenue Boston, MA 02210-1862, USA

#### CONFIDENTIAL

This document contains confidential information. Any use, distribution, or disclosure without the prior written consent of Vertex Pharmaceuticals Incorporated is strictly prohibited except to the extent required under applicable laws or regulations. Persons to whom the information is disclosed must be informed that the information is confidential and may not be further disclosed by them.

#### 2 PROTOCOL SYNOPSIS

Title A Phase 3, Randomized, Double-blind, Controlled Study Evaluating the Efficacy and Safety of

VX-659 Combination Therapy in Subjects With Cystic Fibrosis Who Are Homozygous for the

F508del Mutation (F/F)

**Brief Title** A Phase 3 Study of VX-659 Combination Therapy in CF Subjects Homozygous for F508del

(F/F)

**Clinical Phase** and Clinical **Study Type** 

Phase 3, efficacy and safety

#### **Objectives**

#### Primary Objective

To evaluate the efficacy of VX-659 in triple combination (TC) with tezacaftor (TEZ) and ivacaftor (IVA) in subjects with cystic fibrosis (CF) who are homozygous for the F508del mutation (F/F)

#### **Secondary Objectives**

- To evaluate the safety of VX-659 in TC with TEZ and IVA
- To evaluate the pharmacodynamics (PD) of VX-659 in TC with TEZ and IVA
- To evaluate the pharmacokinetics (PK) of VX-659, TEZ, and IVA when administered in TC

#### **Endpoints Primary Endpoint**

Absolute change in percent predicted forced expiratory volume in 1 second (ppFEV<sub>1</sub>) from baseline at Week 4

#### **Key Secondary Endpoints**

- Absolute change in sweat chloride (SwCl) from baseline at Week 4
- Absolute change in CF Questionnaire-Revised (CFQ-R) respiratory domain score from baseline at Week 4

#### **Other Secondary Endpoints**

- Safety and tolerability assessments based on adverse events (AEs), clinical laboratory values, ECGs, vital signs, and pulse oximetry
- PK parameters of VX-659, TEZ, M1-TEZ, and IVA

Number of Approximately 100 subjects will be randomized (1:1) to the TC VX-659/TEZ/IVA arm or the Subjects TEZ/IVA arm.

**Study** Male and female subjects with CF who are 12 years of age or older who are homozygous for **Population** F508del (F/F)

# Investigational Drug

During the TEZ/IVA Run-in Period, study drug refers to TEZ/IVA and IVA.

During the Treatment Period, study drug refers to VX-659/TEZ/IVA and matching placebo, TEZ/IVA and matching placebo, and IVA.

Active study drugs will be orally administered as fixed-dose combination (FDC) film-coated tablets (2 VX-659/TEZ/IVA tablets or 1 TEZ/IVA tablet) in the morning and as 1 film-coated IVA tablet in the evening.

**Active substance:** VX-659, TEZ (tezacaftor; VX-661), and IVA (ivacaftor; VX-770) **Activity:** CFTR corrector, CFTR corrector, and CFTR potentiator (increased Cl<sup>-</sup> secretion)

Strength: 120 mg/50 mg/75 mg

**Active substance:** TEZ (tezacaftor; VX-661) and IVA (ivacaftor; VX-770) **Activity:** CFTR corrector and CFTR potentiator (increased Cl<sup>-</sup> secretion)

Strength: 100 mg/150 mg

Active substance: IVA (ivacaftor; VX-770)

**Activity:** CFTR potentiator (increased Cl<sup>-</sup> secretion)

Strength: 150 mg

#### **Study Duration**

The total study duration is approximately 16 weeks (4 weeks for the Screening Period, 4 weeks for the TEZ/IVA Run-in Period, 4 weeks for the Treatment Period, and 4 weeks for the Safety Follow-up Period).

#### Study Design

This is a Phase 3, randomized, double-blind, active-controlled, parallel-group, multicenter study.



IVA: ivacaftor; N: number of subjects; TC: triple combination; TEZ: tezacaftor

In the TEZ/IVA Run-in Period, all subjects will receive TEZ 100 mg once daily (qd)/IVA 150 mg every 12 hours (q12h). After completing the TEZ/IVA Run-in Period, subjects will be randomized (1:1) to the TC arm or TEZ/IVA arm for the Treatment Period. The Treatment Period dosages to be evaluated are shown in the table below. Randomization will be stratified by ppFEV<sub>1</sub> determined during the TEZ/IVA Run-in Period (Day -14 assessment; <70 versus  $\geq$ 70) and age at the Screening Visit (<18 versus  $\geq$ 18 years of age). If the Day -14 ppFEV<sub>1</sub> value is not valid or not available, the most recent available ppFEV<sub>1</sub> value will be used for stratification.

#### **Treatment Period Arms and Dosages**

| Treatment Arm | VX-659 Dosage | TEZ Dosage | IVA Dosage |
|---------------|---------------|------------|-------------|
| TC | 240 mg qd | 100 mg qd | 150 mg q12h |
| TEZ/IVA | 0 mg | 100 mg qd | 150 mg q12h |

IVA: ivacaftor; q12h: every 12 hours; qd: once daily; TC: triple combination; TEZ: tezacaftor

**Assessments** Efficacy: Spirometry and CFQ-R

PD: SwCl

Safety: AEs, clinical laboratory assessments, ECGs, vital signs, pulse oximetry, and physical

examinations

PK: VX-659, TEZ, M1-TEZ, and IVA plasma concentrations



The primary efficacy endpoint is the absolute change in ppFEV<sub>1</sub> from baseline at Week 4. The primary null hypothesis to be tested is that the mean absolute change in ppFEV<sub>1</sub> from baseline at Week 4 is the same for the TC and TEZ/IVA treatment groups. The null hypothesis will be tested at a 2-sided significance level of 0.05.

Assuming a within-group SD of 7 percentage points and a 5% dropout rate at Week 4, a sample size of 50 subjects in each treatment group for a total of 100 subjects will have approximately 93% power to detect a difference of 5.0 percentage points for the mean absolute change in ppFEV<sub>1</sub> from baseline at Week 4 between the 2 treatment groups, based on a 2-sided 2-sample *t*-test at a significance level of 0.05.

The primary analysis will be based on a mixed-effects model for repeated measures (MMRM). The model will include the absolute change from baseline in ppFEV<sub>1</sub> at Day 15 and Week 4 as the dependent variable; treatment group, visit, and treatment-by-visit as fixed effects; with continuous baseline ppFEV₁ and age at screening (<18 versus ≥18 years of age) as covariates; and an unstructured covariance structure for the within-subject errors.

The primary result obtained from the model will be the estimated treatment difference at Week 4. The adjusted mean with a 2-sided 95% CI and a 2-sided P value will be provided.

The safety endpoints include AEs, clinical laboratory values, ECGs, vital signs, and pulse oximetry through the Safety Follow-up Visit. The safety analysis will be descriptive only.

#### **IDMC Reviews**

An independent data monitoring committee (IDMC) will conduct safety review of study data as outlined in the IDMC charter.

#### 3 SCHEDULE OF ASSESSMENTS

Table 3-1 and Table 3-2 provide the schedule of assessments for the study.

All visits are to be scheduled relative to the Day 1 Visit (first dose of randomized study drug in the Treatment Period). For example, the Week 4 ( $\pm$  5 days) Visit would occur after 4 weeks of study drug administration in the Treatment Period has been completed.

The Cystic Fibrosis Questionnaire–Revised (CFQ-R),

must be completed before any other assessment at relevant clinic visits. Remaining assessments may be performed in any order when more than 1 assessment is required at a particular time point. All assessments will be performed before study drug dosing (Section 9.6.1), unless noted otherwise.

Table 3-1 Study VX17-659-103: Screening

| Event/Assessment | Screening Period (Day -56 Through Day -29) |
|---|---|
| ICF and assent (when applicable) | X |
| Inclusion and exclusion criteria review | X |
| Demographics | X |
| Medical history | X |
| CFQ-R <sup>a</sup> | X |
| CFTR genotype <sup>b</sup> | X |
| G6PD activity test | X |
| FSH <sup>c</sup> | X |
| Serum pregnancy test (all females of childbearing potential) <sup>d</sup> | X |
| Hematology | X |
| Coagulation | X |
| Serum chemistry | X |
| Urinalysis | X |
| Weight and height <sup>e</sup> | X |
| Ophthalmologic examination <sup>f</sup> | X |
| Complete physical examination | X |
| Vital signs <sup>g</sup> | X |
| Pulse oximetry <sup>g</sup> | X |
| Standard 12-lead ECG <sup>h</sup> | X |
| Spirometry <sup>i</sup> | X |
| Medications review <sup>j</sup> | X |
| Sweat chloride | X |
| AEs and SAEs | Continuous from signing of the ICF through completion of study participation |

AE: adverse events; CFQ-R: CF-Questionnaire-Revised; FSH: follicle-stimulating hormone; G6PD: glucose-6-phosphate dehydrogenase; ICF: informed consent form; SAE: serious adverse event

- <sup>a</sup> The CFQ-R must be completed before the start of any other assessments scheduled for that visit.
- <sup>b</sup> *CFTR* genotyping will be performed for all subjects. If the screening *CFTR* genotype result is not received before Day -28, a previous *CFTR* genotype laboratory report may be used to establish eligibility. Subjects who have been enrolled and whose screening genotype does not confirm study eligibility must be discontinued from the study (Section 9.9).
- FSH will be measured for any suspected postmenopausal female with at least 12 months of continuous spontaneous amenorrhea. Serum FSH levels must be in the postmenopausal range, as determined by the laboratory performing the test, to be considered postmenopausal.
- d Any female subject who does not meet the criteria for non-childbearing potential is considered to be of childbearing potential and must have a serum pregnancy test. A definition of non-childbearing potential is provided in Section 11.7.7.1.
- e Weight and height will be measured with shoes off.
- Ophthalmologic examinations will be conducted only for subjects who are <18 years of age on the date of informed consent. For subjects with documentation of bilateral lens removal, ophthalmologic examinations are not required. The ophthalmologic examination does not need to be conducted if there is documentation of an examination meeting the protocol requirements that was conducted within 3 months before the date of informed consent (Section 11.7.6). The ophthalmologic examination will be conducted by a licensed ophthalmologist or optometrist.
- Vital signs and pulse oximetry will be collected after the subject has been at rest for at least 5 minutes.
- A standard 12-lead ECG will be performed after the subject has been at rest for at least 5 minutes.
- Spirometry may be performed pre- or post-bronchodilator (Section 11.6.1).
- Refer to Section 9.5 for details.

Table 3-2 VX17-659-103: TEZ/IVA Run-in Period, Treatment Period, and Safety Follow-up Visit

| | | Run-in Period<br>Veeks) | Trea | ntment Period (4 V | Veeks) | ETT<br>Visit <sup>b</sup> | Safety Follow-up Visit<br>28 (± 7) Days<br>After the Last Dose of<br>Study Drug (If Applicable) <sup>c</sup> |
|---|---|---|---|---|---|---|---|
| Event/Assessment <sup>a</sup> | Day -28<br>± 1 Day | Day -14<br>(Day -15 to<br>Day -3) | Day 1 <sup>d</sup> | Day 15<br>± 3 Days | Week 4<br>± 5 Days | | |
| Clinic visit | X | X | X | X | X | X | X |
| Inclusion and exclusion criteria confirmation | X | | | | | | |
| CFQ-R <sup>e</sup> | | | X | X | X | X | X |
| Weight and height <sup>f</sup> | X | | X | X | X | X | X |
| Physical examination <sup>g</sup> | Abbreviated | | Complete | | Complete | Complete | |
| Pregnancy testing <sup>h</sup> | Urine | | Urine | | Urine | Serum | Serum |
| Standard 12-lead ECG <sup>i</sup> | X | | X | X | X | X | X |

<sup>&</sup>lt;sup>a</sup> All assessments will be performed before dosing unless noted otherwise.

To enter the Treatment Period, conditions for entry (Section 9.1.3) must be satisfied.

e The CFQ-R, must be completed before any other assessments scheduled at relevant visits. Refer to Section 11.6.2 and

- Weight and height will be measured with shoes off. Following screening, height will be collected only for subjects ≤21 years of age on the date of informed consent.
- Abbreviated and complete physical examinations are defined in Section 11.7.3. Symptom-directed physical examinations will occur at any time during the study if deemed necessary by the investigator.
- Any female subject who does not meet the criteria for non-childbearing potential is considered to be of childbearing potential and must have pregnancy testing at the indicated time points. A definition of non-childbearing potential is provided in Section 11.7.7.1.
- All standard 12-lead ECGs will be performed after the subject has been at rest for at least 5 minutes. ECGs will be collected before dosing (as applicable).

b If the subject prematurely discontinues study drug treatment, an ETT Visit should be scheduled as soon as possible after the decision to discontinue treatment. Subjects who prematurely discontinue treatment during the Treatment Period will continue to complete all scheduled study visits for assessments following completion of the ETT Visit (Section 9.1.5.2).

The Safety Follow-Up Visit is required for all subjects, unless the subject completes the Week 4 Visit and has enrolled in a separate open-label study within 28 days after the last dose of study drug (Section 9.1.4). If an ETT Visit occurs 3 weeks or later following the last dose of study drug, then the ETT Visit replaces the Safety Follow-up Visit (Section 9.1.5).

Table 3-2 VX17-659-103: TEZ/IVA Run-in Period, Treatment Period, and Safety Follow-up Visit

| | | Run-in Period<br>Weeks) | Trea | atment Period (4 V | Veeks) | ETT<br>Visit <sup>b</sup> | Safety Follow-up Visit 28 (± 7) Days After the Last Dose of Study Drug (If Applicable) <sup>c</sup> |
|---|---|---|---|---|---|---|---|
| Event/Assessment <sup>a</sup> | Day -28<br>± 1 Day | Day -14<br>(Day -15 to<br>Day -3) | Day 1 <sup>d</sup> | Day 15<br>± 3 Days | Week 4<br>± 5 Days | | |
| Vital signs <sup>j</sup> | X | | X | X | X | X | X |
| Pulse oximetry <sup>j</sup> | X | | X | X | X | X | X |
| Spirometry <sup>k</sup> | | X | X | X | X | X | X |
| Sweat chloride <sup>1</sup> | | X | X | X | X | X | |
| Urinalysis | X | | X | | X | X | X |
| Hematology | X <sup>m</sup> | | X <sup>m</sup> | X | X | X | X |
| Coagulation | X <sup>m</sup> | | X <sup>m</sup> | | X | X | X |
| Serum chemistry | X <sup>m</sup> | | X <sup>m</sup> | X | X | X | X |
| PK sampling <sup>n</sup> | | | X | | X | X | |

Vital signs and pulse oximetry will be collected before dosing and after the subject has been at rest for at least 5 minutes.

Spirometry assessments must be performed before study drug dosing (see Section 9.6.1) and should be performed pre-bronchodilator (Section 11.6.1) at approximately the same time at each visit.

Sweat chloride collection will occur before study drug dosing (Section 11.4). At each time point, 2 samples will be collected, 1 from each arm (left and right).

<sup>&</sup>lt;sup>m</sup> Blood samples will be collected before the first dose of study drug in each study period.

The Day 1 predose PK sample must be collected before dosing. The Week 4 predose PK sample must be collected within 60 minutes before dosing for subjects who are receiving their first dose of study drug in an open-label study on the same day as the Week 4 Visit. For subjects who are not entering an open-label study on the same day as the Week 4 Visit the Week 4 Visit (Section 11 3 1)

Table 3-2 VX17-659-103: TEZ/IVA Run-in Period, Treatment Period, and Safety Follow-up Visit

| | | Run-in Period<br>Veeks) | Trea | ntment Period (4 V | Veeks) | ETT<br>Visit <sup>b</sup> | Safety Follow-up Visit 28 (± 7) Days After the Last Dose of Study Drug (If Applicable) <sup>c</sup> |
|---|---|---|---|---|---|---|---|
| Event/Assessment <sup>a</sup> | Day -28<br>± 1 Day | Day -14<br>(Day -15 to<br>Day -3) | Day 1 <sup>d</sup> | Day 15<br>± 3 Days | Week 4<br>± 5 Days | | |
| Run-in TEZ/IVA dosing <sup>q</sup> | Day -28 to eve | ening on Day -1 | | | | | |
| Run-in TEZ/IVA drug count | X | X | X | | | | |
| Randomization <sup>r</sup> | | | X | | | | |
| Randomized study drug dosing <sup>s</sup> | | | Day 1 throug | h evening before th | e Week 4 Visit | | |
| Randomized study drug count | | | X | X | X | X | |
| Medications review <sup>u</sup> | | Co | ontinuous from s | igning of ICF throu | igh completion of | study participatio | n |
| Treatments and procedures review <sup>u</sup> | | Co | ontinuous from s | igning of ICF throu | igh completion of | study participatio | n |
| AEs and SAEs <sup>u, v</sup> | | Co | ontinuous from s | igning of ICF throu | igh completion of | study participatio | n |

AE: adverse event; CF: cystic fibrosis; CFQ-R: CF Questionnaire-Revised; ETT: Early Termination of Treatment; GPS: Global Patient Safety; ICF: informed consent form; IV: intravenous; IVA: ivacaftor; PD: pharmacodynamic; PK: pharmacokinetic; SAE: serious adverse event; TEZ: tezacaftor;

Completion of study participation is defined in Section 9.1.7.

<sup>&</sup>lt;sup>q</sup> For the Run-in Period, TEZ/IVA should be administered as outlined in Section 9.6.1. On days of scheduled visits, refer to Section 9.6.1 for the timing of dosing relative to the assessments. The final dose during the Run-in Period will be administered on Day -1, the evening before the Day 1 Visit.

Randomization may occur on either Day -1 or Day 1, after conditions for entry into the Treatment Period (Section 9.1.3) have been satisfied. Randomization must occur before the first dose of study drug in the Treatment Period.

For the Treatment Period, the randomized study drug regimen should be administered as outlined in Section 9.6.1. On days of scheduled visits, refer to Section 9.6.1 for the timing of dosing relative to the assessments. The final dose of study drug in the Treatment Period will be administered the evening before the Week 4 Visit.

SAEs that occur after completion of study participation and are considered related to study drug will be reported to Vertex GPS within 24 hours as described in Section 13.1.2.2.

## 4 TABLE OF CONTENTS

| 1 | Title Page | 1 |
|------------|--------------------------------------------------------|----|
| • | | |
| 2 | v 1 | |
| <b>3 4</b> | | |
| 4 | Table of Contents List of Tables | |
| | List of Figures | |
| | List of Abbreviations. | |
| 5 | | |
| J | 5.1 Background | |
| | 5.2 Rationale for the Present Study | |
| 6 | | |
| | 6.1 Primary Objective | |
| | 6.2 Secondary Objectives | |
| 7 | | |
| | 7.1 Primary Endpoint | |
| | 7.2 Secondary Endpoints | 20 |
| | 7.2.1 Key Secondary Endpoints | 20 |
| | 7.2.2 Other Secondary Endpoints | 20 |
| 8 | · I | |
| | 8.1 Inclusion Criteria | |
| _ | 8.2 Exclusion Criteria | |
| 9 | $oldsymbol{v}$ | |
| | 9.1 Study Design 9.1.1 Screening | |
| | 9.1.1 Screening | |
| | 9.1.1.1 Repetition of Screening Assessment(s) | |
| | 9.1.1.2 Rescreening Period Window | |
| | 9.1.2 Tezacaftor/Ivacaftor Run-in Period | |
| | 9.1.3 Treatment Period | |
| | 9.1.4 Follow-up. | |
| | 9.1.5 Early Termination of Treatment | 25 |
| | 9.1.5.1 Discontinuation During the Run-in Period | |
| | 9.1.5.2 Discontinuation During the Treatment Period | |
| | 9.1.6 Lost to Follow-up | |
| | 9.1.7 Completion of Study Participation | 26 |
| | 9.1.8 Independent Data Monitoring Committee | |
| | 9.2 Method of Assigning Subjects to Treatment Groups | |
| | 9.3 Rationale for Study Design and Study Drug Regimens | |
| | 9.3.1 Study Design | |
| | 9.3.2 Study Drug Dose | |
| | 9.3.3 Rationale for Study Population | |
| | 9.3.4 Rationale for Study Assessments | 28 |

| 9.4.2 Ex<br>9.5 Prior ar<br>9.6 Admini<br>9.6.1 Do<br>9.6.2 M<br>9.6.2.1<br>9.6.2.2<br>9.7 Dose M<br>9.8 Study I<br>9.8.1 Li<br>9.8.2 Ra<br>9.9 Remov<br>9.10 Replace<br>10 Study Drug<br>10.1 Prepara | Exposure to Sunlight 30 for and Concomitant Medications 30 Iministration 3 Dosing 3 Missed Doses 3 2.1 Morning Dose of Study Drug 3 2.2 Evening Dose of Study Drug 3 Ose Modification for Toxicity 3 ady Drug Interruption and Stopping Rules 3 | 0<br>0<br>1<br>1<br>2<br>2<br>2<br>2<br>2<br>3 |
|---|---|---|
| 9.5 Prior and 9.6 Administration 9.6.1 Do 9.6.2 M 9.6.2.1 9.6.2.2 9.7 Dose M 9.8 Study I 9.8.1 Lings 9.8.2 Ray 9.9 Remove 9.10 Replace 10 Study Drug 10.1 Prepara | for and Concomitant Medications36lministration3Dosing3Missed Doses362.1 Morning Dose of Study Drug362.2 Evening Dose of Study Drug36ose Modification for Toxicity36ody Drug Interruption and Stopping Rules36Liver Function Tests36Rash36moval of Subjects36placement of Subjects36 | 0<br>1<br>1<br>2<br>2<br>2<br>2<br>2<br>3 |
| 9.6 Admini<br>9.6.1 Do<br>9.6.2 M<br>9.6.2.1<br>9.6.2.2<br>9.7 Dose M<br>9.8 Study I<br>9.8.1 Li<br>9.8.2 Ra<br>9.9 Remov<br>9.10 Replace<br>10 Study Drug<br>10.1 Prepara | Iministration3Dosing3Missed Doses32.1 Morning Dose of Study Drug32.2 Evening Dose of Study Drug3Ose Modification for Toxicity3Idy Drug Interruption and Stopping Rules3Liver Function Tests3Rash3moval of Subjects3placement of Subjects3 | 1<br>1<br>2<br>2<br>2<br>2<br>2<br>3<br>3 |
| 9.6 Admini<br>9.6.1 Do<br>9.6.2 M<br>9.6.2.1<br>9.6.2.2<br>9.7 Dose M<br>9.8 Study I<br>9.8.1 Li<br>9.8.2 Ra<br>9.9 Remov<br>9.10 Replace<br>10 Study Drug<br>10.1 Prepara | Iministration3Dosing3Missed Doses32.1 Morning Dose of Study Drug32.2 Evening Dose of Study Drug3Ose Modification for Toxicity3Idy Drug Interruption and Stopping Rules3Liver Function Tests3Rash3moval of Subjects3placement of Subjects3 | 1<br>1<br>2<br>2<br>2<br>2<br>2<br>3<br>3 |
| 9.6.1 Do 9.6.2 M 9.6.2.1 9.6.2.2 9.7 Dose M 9.8 Study I 9.8.1 Li 9.8.2 Ra 9.9 Remov 9.10 Replace 10 Study Drug 10.1 Prepara | Dosing3Missed Doses32.1 Morning Dose of Study Drug32.2 Evening Dose of Study Drug3ose Modification for Toxicity3ody Drug Interruption and Stopping Rules3Liver Function Tests3Rash3moval of Subjects3placement of Subjects3 | 1<br>2<br>2<br>2<br>2<br>2<br>2<br>3<br>3 |
| 9.6.2 M 9.6.2.1 9.6.2.2 9.7 Dose M 9.8 Study I 9.8.1 Li 9.8.2 Ra 9.9 Remov 9.10 Replace 10 Study Drug 10.1 Prepara | Missed Doses 32 2.1 Morning Dose of Study Drug 33 2.2 Evening Dose of Study Drug 33 2.3 Evening Dose of Study Drug 33 2.4 Evening Dose of Study Drug 33 2.5 Evening Dose of Study Drug 33 2.6 Evening Dose of Study Drug 33 2.7 Evening Dose of Study Drug 33 2.8 Modification for Toxicity 33 2.8 Liver Function and Stopping Rules 33 2.8 Evening Dose of Study Drug 33 2.8 Evening Dose of Study Drug 33 2.9 Evening Dose of Study Drug 33 2.0 Evening Dose of Study Drug 33 2.0 Evening Dose of Study Drug 33 2.1 Evening Dose of Study Drug 33 2.2 Evening Dose of Study Drug 33 2.3 Evening Dose of Study Drug 33 2.4 Evening Dose of Study Drug 33 2.5 Evening Dose of Study Drug 33 2.7 Evening Dose of Study Drug 33 2.8 Evening Dose of Study Drug 33 2.8 Evening Dose of Study Drug 34 2.8 Evening Dose o | 2<br>2<br>2<br>2<br>2<br>2<br>3<br>3 |
| 9.6.2.1<br>9.6.2.2<br>9.7 Dose M<br>9.8 Study I<br>9.8.1 Li<br>9.8.2 Ra<br>9.9 Remov<br>9.10 Replace<br>10 Study Drug<br>10.1 Prepara | 2.1 Morning Dose of Study Drug362.2 Evening Dose of Study Drug37Ose Modification for Toxicity36Idy Drug Interruption and Stopping Rules37Liver Function Tests37Rash38moval of Subjects38placement of Subjects38 | 2<br>2<br>2<br>2<br>3<br>3 |
| 9.6.2.2 9.7 Dose M 9.8 Study I 9.8.1 Li 9.8.2 Ra 9.9 Remov 9.10 Replace 10 Study Drug 10.1 Prepara | 2.2 Evening Dose of Study Drug | 2<br>2<br>2<br>2<br>3<br>3 |
| 9.7 Dose M<br>9.8 Study I<br>9.8.1 Li<br>9.8.2 Ra<br>9.9 Remov<br>9.10 Replace<br>10 Study Drug<br>10.1 Prepara | ose Modification for Toxicity | 2<br>2<br>2<br>3<br>3 |
| 9.8 Study I<br>9.8.1 Li<br>9.8.2 Ra<br>9.9 Remov<br>9.10 Replace<br>10 Study Drug<br>10.1 Prepara | Idy Drug Interruption and Stopping Rules33Liver Function Tests33Rash33moval of Subjects33placement of Subjects34 | 2 3 3 |
| 9.8.1 Li<br>9.8.2 Ra<br>9.9 Remov<br>9.10 Replace<br>10 Study Drug<br>10.1 Prepara | Liver Function Tests 3 Rash 3 moval of Subjects 3 placement of Subjects 3 | 2 3 3 |
| 9.8.2 Ra<br>9.9 Remov<br>9.10 Replace<br>10 <b>Study Drug</b><br>10.1 Prepara | Rash 33 moval of Subjects 35 placement of Subjects 36 | 3 |
| 9.9 Remov<br>9.10 Replace<br>10 Study Drug<br>10.1 Prepara | moval of Subjects 3. placement of Subjects 3. | 3 |
| 9.10 Replace<br>10 Study Drug<br>10.1 Prepara | placement of Subjects | |
| 10 Study Drug<br>10.1 Prepara | | + |
| 10.1 Prepara | Drug information and Management | |
| • | eparation and Dispensing 34 | |
| то д Раскар | ckaging and Labeling 3 | |
| | idy Drug Supply, Storage, and Handling | |
| | ug Accountability | |
| | sposal, Return, or Retention of Unused Drug | |
| | • | |
| | inding and Unblinding 30 | |
| | Blinding 30 | |
| | Unblinding 3 | |
| | ments | |
| _ | ming of Assessments. | |
| | bject and Disease Characteristics | |
| | armacokinetics | |
| 11.4 Pharma | armacodynamics: Sweat Chloride | 9 |

| | 11.7 Safety | | 42 |
|---|---|---|---|
| | 11.7.1 Adverse Events | | 43 |
| | 11.7.2 Clinical Laboratory As | ssessments | 43 |
| | 11.7.3 Physical Examinations | and Vital Signs | 44 |
| | 11.7.4 Pulse Oximetry | | 45 |
| | 11.7.5 Electrocardiograms | | 45 |
| | 11.7.6 Ophthalmologic Exam | ination | 45 |
| | 11.7.7 Contraception and Pre | gnancy4 | 46 |
| | 11.7.7.1 Contraception | | 46 |
| | 11.7.7.2 Pregnancy | | 47 |
| <b>12</b> | 12 Statistical and Analytical Plan | S | <b>48</b> |
| | 12.1 Sample Size and Power | | 48 |
| | 12.2 Analysis Sets | | 48 |
| | 12.3.1 General Consideration | S | 48 |
| | 12.3.2 Background Character | istics | 49 |
| | 12.3.2.1 Subject Dispositio | n ' | 49 |
| | | Baseline Characteristics | |
| | | itant Medications | |
| | 12.3.2.4 Study Drug Expos | ure and Compliance | 50 |
| | | Deviations | |
| | | odynamic Analyses | |
| | 12.3.3.1 Analysis of Primar | y Variable | 51 |
| | 12.3.3.2 Analysis of Key S | econdary Variables | 51 |
| | | tment | |
| | | y Assessments | |
| | 5 | | |
| | | ion | |
| | 12.3.4.7 Other Safety Anal | ysis | 54 |
| | | alyses | |
| | <u> - </u> | | |
| | | lysis | |
| | | ysis | |
| 13 | | ry, and Administrative Considerations | <b>55</b> |
| | | Adverse Event Documentation, Severity Grading, and | |
| | 1 0 | | |
| | | dverse Event | |
| | 13.1.1.2 Clinically Signific | ant Assessments | 55 |

| 13.1.1.3 Documentation of Adverse Events | 56 |
|--------------------------------------------------------------|----|
| 13.1.1.4 Adverse Event Severity | 56 |
| 13.1.1.5 Adverse Event Causality | 56 |
| 13.1.1.6 Study Drug Action Taken | 57 |
| 13.1.1.7 Adverse Event Outcome | 57 |
| 13.1.1.8 Treatment Given | 58 |
| 13.1.2 Serious Adverse Events | 58 |
| 13.1.2.1 Definition of a Serious Adverse Event | 58 |
| 13.1.2.2 Documentation of Serious Adverse Events | 59 |
| 13.1.2.3 Reporting Serious Adverse Events | 59 |
| 13.1.2.4 Expedited Reporting and Investigator Safety Letters | 59 |
| 13.2 Administrative Requirements | |
| 13.2.1 Ethical Considerations | 60 |
| 13.2.2 Subject Information and Informed Consent | 60 |
| 13.2.3 Investigator Compliance | 60 |
| 13.2.4 Access to Records | 60 |
| 13.2.5 Subject Privacy | 60 |
| 13.2.6 Record Retention | 61 |
| 13.2.7 Study Termination | 61 |
| 13.2.8 End of Study | 61 |
| 13.3 Data Quality Assurance | 62 |
| 13.4 Monitoring | |
| 13.5 Electronic Data Capture | 62 |
| 13.6 Publications and Clinical Study Report | 63 |
| 13.6.2 Clinical Study Report | 63 |
| 14 References | 64 |
| 15 Protocol Signature Pages | |
| 15.1 Sponsor Signature Page | |
| 15.2 Investigator Signature Page | 67 |

## **List of Tables**

| Table 3-1 | Study VX17-659-103: Screening | 7 |
|---|---|---|
| Table 3-2 | VX17-659-103: TEZ/IVA Run-in Period, Treatment Period, and Safety | |
| | Follow-up Visit | 8 |
| Table 9-1 | Treatment Period Arms and Dosages | |
| Table 9-2 | Prohibited Medications | 30 |
| Table 10-1 | Study Drug: Strength/Dosing Form/Route | 35 |
| Table 11-1 | Safety Laboratory Test Panels | 43 |
| Table 11-2 | Acceptable Methods of Contraception | 47 |
| Table 13-1 | Grading of AE Severity | 56 |
| Table 13-2 | Classifications for AE Causality | 57 |
| Table 13-3 | Classifications for Study Drug Action Taken With Regard to an AE | 57 |
| Table 13-4 | Classifications for Outcome of an AE | |
| List of Figu | ıres | |
| Figure 9-1 | Schematic of the Study Design | 23 |

## **List of Abbreviations**

| Abbreviation | Term |
|---|---|
| AE | adverse event |
| ALP | alkaline phosphatase |
| ALT | alanine transaminase |
| AST | aspartate transaminase |
| CBC | complete blood count |
| CF | cystic fibrosis |
| CFQ-R | Cystic Fibrosis Questionnaire-Revised |
| CFTR | CF transmembrane conductance regulator gene |
| CFTR | CF transmembrane conductance regulator protein |
| Cl <sup>-</sup> | chloride ion |
| CPAP | clinical pharmacology analysis plan |
| CRF | case report form |
| CRO | contract research organization |
| CSR | clinical study report |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CYP | cytochrome P450 |
| ECG | electrocardiogram |
| EDC | electronic data capture |
| EENT | eyes, ears, nose, and throat |
| ETT | Early Termination of Treatment |
| EU | European Union |
| F508del | CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein |
| F/F | homozygous for F508del |
| F/MF | heterozygous for F508del and a minimal CFTR function mutation |
| FAS | Full Analysis Set |
| FDA | Food and Drug Administration |
| FDC | fixed-dose combination |
| $FEV_1$ | forced expiratory volume in 1 second |
| FSH | follicle-stimulating hormone |
| G551D | |
| G551D | CFTR missense gene mutation that results in the replacement of a glycine residue at position 551 of CFTR with an aspartic acid residue |
| G6PD | Glucose-6-phosphate dehydrogenase |
| GCP | Good Clinical Practice |
| GGT | gamma-glutamyl transferase |
| GLI | Global Lung Function Initiative |
| GPS | Global Patient Safety |
| HIPAA | Health Insurance Portability and Accountability Act |
| HR | heart rate |
| ICF | informed consent form |
| ICH | International Council for Harmonization |

| Abbreviation | Term |
|---|---|
| IDMC | independent data monitoring committee |
| IEC | independent ethics committee |
| IPD | important protocol deviation |
| IRB | institutional review board |
| IV | intravenous |
| IVA | ivacaftor |
| IWRS | interactive web response system |
| LLN | lower limit of normal |
| LUM | lumacaftor |
| M1-TEZ | metabolite of TEZ |
| MAA | Marketing Authorization Application |
| max | maximum value |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MF | minimal CFTR function mutation |
| min | minimum value |
| MMRM | mixed-effects model for repeated measures |
| n | number of subjects |
| OATP1B1 | organic anion transporting polypeptide 1B1 |
| P | probability |
| PD | pharmacodynamic, pharmacodynamics |
| PE | physical examination |
| PEx | pulmonary exacerbation(s) |
| PK | pharmacokinetic, pharmacokinetics |
| $ppFEV_1$ | percent predicted forced expiratory volume in 1 second |
| PR | PR interval, segment |
| PT | Preferred Term |
| q12h | every 12 hours |
| qd | once daily |
| QRS | the portion of an ECG comprising the Q, R, and S waves, together representing ventricular depolarization |
| QT | QT interval |
| QTc | QT interval corrected |
| QTcF | QT interval corrected by Fridericia's formula |
| RR | interval from the onset of 1 QRS complex to the next |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SD | standard deviation |
| SE | standard error |
| SI | SI units (International System of Units) |
| SOC | System Organ Class |
| SUSAR | suspected, unexpected, serious adverse reaction |
| SwCl | sweat chloride |
| TC | triple combination |
| TE | treatment-emergent |
| TEAE | treatment-emergent adverse event |

| Abbreviation | Term |
|--------------|--------------------------|
| TEZ | tezacaftor |
| ULN | upper limit of normal |
| US | United States |
| USA | United States of America |
| UV | ultraviolet |

#### 5 INTRODUCTION

## 5.1 Background

Cystic fibrosis (CF) is an autosomal recessive chronic disease with serious morbidities and frequent premature mortality. At present, there is no cure. CF affects approximately 70,000 individuals worldwide<sup>1</sup> (approximately 30,000 in the US<sup>1, 2</sup> and 39,000 in the EU<sup>3</sup>). Based on its prevalence, CF qualifies as an orphan disease.<sup>4, 5</sup>

CF is caused by decreased quantity and/or function of the CFTR protein due to mutations in the *CFTR* gene. The CFTR protein is an epithelial chloride channel that aids in regulating salt and water absorption and secretion and pH balance in sweat glands and multiple organs, including the lungs, pancreas, and other gastrointestinal organs. Despite progress in the treatment of CF with antibiotics and mucolytics, the predicted median age of survival for a person with CF is approximately 40 years.<sup>2,6</sup> Progressive loss of lung function is the leading cause of mortality.<sup>7</sup> More effective treatments are needed for CF.

The most common disease-causing *CFTR* mutation, *F508del*, accounts for 70% of the identified alleles in people with  $CF^8$ , and approximately 40% of people with CF are homozygous for *F508del* (F/F).<sup>2, 3, 8</sup>

Based on the understanding of the molecular defects caused by *CFTR* mutations, 2 complementary approaches have been developed to address the decreased quantity and/or function of CFTR in order to enhance chloride transport in patients with CF. Correctors facilitate the cellular processing and trafficking to increase the quantity of functional CFTR at the cell surface. Potentiators increase the channel open probability of the CFTR protein delivered to the cell surface to enhance ion transport. Depending on the amount of residual CFTR channel activity in the membrane, and the pathophysiology of that activity (reflecting the *CFTR* genotype of the patient and possibly other factors), both approaches may be required.

The therapeutic activity of CFTR correctors and potentiators has been established with products that were developed by Vertex and approved for the treatment of CF: ivacaftor (IVA) monotherapy (Kalydeco<sup>®</sup>), and lumacaftor (LUM) in combination with IVA (Orkambi<sup>®</sup>). Kalydeco and Orkambi are approved to treat CF in patients with specific *CFTR* genotypes. A second corrector/potentiator combination, tezacaftor (TEZ)/IVA (Symdeko®) is now approved in the US. An MAA has been submitted and is under review.

VX-659 is a next-generation CFTR corrector being developed for administration in triple combination (TC) with TEZ/IVA for the treatment of CF.

## 5.2 Rationale for the Present Study

This study will evaluate the efficacy and safety of VX-659 in TC with TEZ/IVA in subjects with CF who have an F/F genotype. These patients have continuing unmet need despite currently available CFTR modulators. The potential for benefit in these patients is supported by in vitro data and clinical data in subjects with a single responsive *F508del* allele; in addition, the TC of VX-659/TEZ/IVA is generally safe and well tolerated (refer to VX-659 Investigator's Brochure).

#### 6 STUDY OBJECTIVES

## 6.1 Primary Objective

To evaluate the efficacy of VX-659 in TC with TEZ and IVA in subjects with CF who are homozygous for the *F508del* mutation (F/F)

## 6.2 Secondary Objectives

- To evaluate the safety of VX-659 in TC with TEZ and IVA
- To evaluate the pharmacodynamics (PD) of VX-659 in TC with TEZ and IVA
- To evaluate the pharmacokinetics (PK) of VX-659, TEZ, and IVA when administered in TC

#### 7 STUDY ENDPOINTS

## 7.1 Primary Endpoint

Absolute change in ppFEV<sub>1</sub> from baseline at Week 4

## 7.2 Secondary Endpoints

## 7.2.1 Key Secondary Endpoints

- Absolute change in sweat chloride (SwCl) from baseline at Week 4
- Absolute change in CFQ-R respiratory domain score from baseline at Week 4

## 7.2.2 Other Secondary Endpoints

- Safety and tolerability assessments based on adverse events (AEs), clinical laboratory values, ECGs, vital signs, and pulse oximetry
- PK parameters of VX-659, TEZ, M1-TEZ, and IVA



#### 8 STUDY POPULATION

Eligibility will be reviewed and documented by an appropriately qualified member of the investigator's team before subjects receive study drug on Day -28.

Subjects who meet all of the inclusion criteria and none of the exclusion criteria will be eligible.

#### 8.1 Inclusion Criteria

- 1. Subject (or his or her legally appointed and authorized representative) will sign and date an informed consent form (ICF), and, when appropriate, an assent form.
- 2. Willing and able to comply with scheduled visits, treatment plan, study restrictions, laboratory tests, contraceptive guidelines, and other study procedures.

- 3. Age 12 years or older, on the date of informed consent.
- 4. Confirmed diagnosis of CF as determined by the investigator.
- 5. Subject has the F/F genotype. Note: If the screening *CFTR* genotype result is not received before Day -28, a previous *CFTR* genotype laboratory report may be used to establish eligibility. Subjects who have been enrolled and whose screening genotype is not confirmed to be F/F must be discontinued from the study (Section 9.9).
- 6. Forced expiratory volume in 1 second (FEV₁) value ≥40% and ≤90% of predicted mean for age, sex, and height (equations of the Global Lung Function Initiative [GLI])<sup>9</sup> at the Screening Visit. Spirometry measurements must meet American Thoracic Society/European Respiratory Society criteria <sup>10</sup> for acceptability and repeatability.
- 7. Stable CF disease as judged by the investigator.
- 8. Willing to remain on a stable CF treatment regimen (as defined in Section 9.5) through completion of study participation.

#### 8.2 Exclusion Criteria

- 1. History of any illness or any clinical condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug(s) to the subject. This includes, but is not limited to, the following:
  - Clinically significant cirrhosis with or without portal hypertension.
  - Solid organ or hematological transplantation.
  - Alcohol or drug abuse in the past year, including, but not limited to, cannabis, cocaine, and opiates, as deemed by the investigator.
  - Cancer, except for squamous cell skin cancer, basal cell skin cancer, and Stage 0 cervical carcinoma in situ (all 3 with no recurrence for the last 5 years).
- 2. Any of the following abnormal laboratory values at screening:
  - Hemoglobin <10 g/dL
  - Total bilirubin >2 × ULN
  - Aspartate transaminase (AST), alanine transaminase (ALT), gamma-glutamyl transferase (GGT), or alkaline phosphatase (ALP) ≥3 × ULN
  - Abnormal renal function defined as glomerular filtration rate ≤50 mL/min/1.73 m<sup>2</sup> (calculated by the Modification of Diet in Renal Disease Study Equation)<sup>11, 12</sup> for subjects ≥18 years of age and ≤45 mL/min/1.73 m<sup>2</sup> (calculated by the Counahan-Barratt equation)<sup>13</sup> for subjects aged 12 to 17 years (inclusive)
- 3. An acute upper or lower respiratory infection, pulmonary exacerbation(s) (PEx), or changes in therapy (including antibiotics) for sinopulmonary disease within 28 days before the first dose of TEZ/IVA in the Run-in Period (Day -28).
- 4. Lung infection with organisms associated with a more rapid decline in pulmonary status (including, but not limited to, *Burkholderia cenocepacia*, *Burkholderia dolosa*, and *Mycobacterium abscessus*). For subjects who have had a history of a positive culture, the

investigator will apply the following criteria to establish whether the subject is free of infection with such organisms:

- The subject has not had a respiratory tract culture positive for these organisms within the 12 months before the date of informed consent.
- The subject has had at least 2 respiratory tract cultures negative for such organisms within the 12 months before the date of informed consent, with the first and last of these separated by at least 3 months, and the most recent one within the 6 months before the date of informed consent.
- 5. An acute illness not related to CF (e.g., gastroenteritis) within 14 days before the first dose of TEZ/IVA in the Run-in Period (Day -28).
- 6. Ongoing or prior participation in a study of an investigational treatment other than a Vertex CFTR modulator within 28 days or 5 terminal half-lives (whichever is longer) before screening. The duration of the elapsed time may be longer if required by local regulations.
- 7. Use of prohibited medications as defined in Table 9-2, within the specified window before the first dose of TEZ/IVA in the Run-in Period (Day -28).
- 8. Pregnant or nursing females. Females of childbearing potential must have a negative pregnancy test at Screening/Day -56 (serum test) and TEZ/IVA Run-in Period/Day -28 (urine test).
- 9. The subject or a close relative of the subject is the investigator or a subinvestigator, research assistant, pharmacist, study coordinator, or other staff directly involved with the conduct of the study at that site. However, an adult (aged 18 years or older) who is a relative of a study staff member may be enrolled in the study provided that
  - the adult lives independently of and does not reside with the study staff member, and
  - the adult participates in the study at a site other than the site at which the family member is employed.

#### 9 STUDY IMPLEMENTATION

## 9.1 Study Design

This is a Phase 3, randomized, double-blind, active-controlled, parallel-group, multicenter study. A schematic of the study design is shown in Figure 9-1.

**Treatment Period** Screening TEZ/IVA Run-in TC Arm: Safety Follow-up Period Period VX-659/TEZ/IVA N = 50TEZ/IVA Arm: Placebo + TEZ/IVA N = 50 Day -28 to Day -1 28 days Day -56 to Day -29 4 Weeks (Day 1 to Week 4) Open-label Study Day -1 or Day 1 Randomization

Figure 9-1 Schematic of the Study Design

IVA: ivacaftor; N: number of subjects; TC: triple combination; TEZ: tezacaftor

Note: The Safety Follow-up Visit is not required for subjects who complete the Week 4 Visit and have enrolled in an open-label study within 28 days after the last dose of study drug (Section 9.1.4).

Study drug is defined in Section 10.

All subjects entering the TEZ/IVA Run-in Period will receive TEZ 100 mg once daily (qd)/IVA 150 mg every 12 hours (q12h). Following completion of the TEZ/IVA Run-in Period, approximately 100 subjects will be randomized (1:1) to the TC arm or TEZ/IVA arm for the Treatment Period. The planned dosages for the Treatment Period are shown in Table 9-1. Randomization will be stratified; details are provided in Section 9.2.

Table 9-1 Treatment Period Arms and Dosages

| Treatment Arm | VX-659 Dosage | TEZ Dosage | IVA Dosage |
|---------------|---------------|------------|-------------|
| TC | 240 mg qd | 100 mg qd | 150 mg q12h |
| TEZ/IVA | 0 mg | 100 mg qd | 150 mg q12h |

IVA: ivacaftor; q12h: every 12 hours; qd: once daily; TC: triple combination; TEZ: tezacaftor Note: Study drug administration is described in Section 9.6.

Study visits and assessments to be conducted are shown in Table 3-1 and Table 3-2. All visits will occur within the windows specified.

#### 9.1.1 Screening

The Screening Period (Day -56 through Day -29) will occur within 28 days before the first dose of study drug in the Run-in Period.

Screening assessments will be used to confirm that subjects meet the eligibility criteria. The investigator (or an appropriate authorized designee) will obtain informed consent and assent, if applicable, from each subject before any study procedure takes place.

## 9.1.1.1 Repetition of Screening Assessment(s)

Screening assessments may be repeated once to establish study eligibility. If repeat values of the individual assessment(s) are within the eligibility criteria and completed within the screening window, then the subject is eligible for the study.

#### 9.1.1.2 Rescreening

Subjects may be rescreened once. If a subject is rescreened, all screening assessments will be repeated, except for:

- *CFTR* genotyping
- Follicle-stimulating hormone (FSH) level (if serum FSH level was in the postmenopausal range as determined by the laboratory performing the test during prior screening)
- G6PD activity test
- Ophthalmologic examination (if performed within 3 months of the date of informed consent, for subjects <18 years of age)

If a subject is rescreened, a new screening window will begin when the first rescreening assessment has been initiated.

#### 9.1.1.3 Extension of Screening Period Window

A subject may have the Screening Period window extended by 2 weeks for the following reasons:

- Repetition of the Screening Period assessments (Section 9.1.1.1)
- Unexpected operational or logistic delays, or to meet the eligibility criteria
- Scheduling of ophthalmologic examination (for subjects <18 years of age on the date of informed consent, Section 11.7.6)

#### 9.1.2 Tezacaftor/Ivacaftor Run-in Period

The TEZ/IVA Run-in Period has a 4-week duration and is designed to establish a reliable on-treatment (TEZ/IVA) baseline for the Treatment Period. The first dose of open-label TEZ/IVA will be administered at the Day -28 Visit. The last dose of open-label TEZ/IVA will be administered in the evening on Day -1 (1 day before the Day 1 Visit).

On Day -14, spirometry and SwCl will be assessed. The Day -14 spirometry assessment will be used for stratification of randomization (Section 9.2).

Subjects who prematurely discontinue study drug treatment during the Run-in Period will not be randomized or participate in the Treatment Period (Section 9.1.5.1).

#### 9.1.3 Treatment Period

The Treatment Period will be randomized, double-blind, and active-controlled. It will last approximately 4 weeks (Day 1 to Week 4). Study drug administration details are provided in Section 9.6

Randomization will occur before the first dose of study drug during the Treatment Period and may occur on either Day -1 or Day 1. Randomization and stratification details are provided in Section 9.2

To enter the Treatment Period, subjects must have stable CF disease (as judged by the investigator) and have remained on a stable CF treatment regimen during the TEZ/IVA Run-in Period. Female subjects of childbearing potential also must have a negative pregnancy test at Day 1 before receiving randomized study drug. If these conditions are not met (for example, if the subject has an acute upper or lower respiratory infection, PEx, or changes in therapy [including antibiotics] for sinopulmonary disease within 28 days before the Day 1 Visit [first dose of study drug in the Treatment Period]), subjects may be rescreened once (Section 9.1.1.2) and re-enter the Run-in Period on Day -28.

Subjects who prematurely discontinue study drug treatment during the Treatment Period will remain in the study from the time of discontinuation of study drug treatment through the last scheduled study visit and complete the assessments for all study visits, as described in Section 9.1.5.2.

#### 9.1.4 Follow-up

The Safety Follow-up Visit will occur approximately 28 days after the last dose of study drug for subjects who complete study drug dosing and for subjects who prematurely discontinue study drug dosing, as described in Section 9.1.5.

An open-label study will be available for subjects who complete the Week 4 Visit and are eligible. The Safety Follow-up Visit is not required for subjects who complete the Week 4 Visit and enroll in an open-label study within 28 days after the last dose of study drug.

#### 9.1.5 Early Termination of Treatment

If a subject prematurely discontinues study drug treatment, an Early Termination of Treatment (ETT) Visit should be scheduled as soon as possible after the decision to discontinue treatment. Subjects who prematurely discontinue treatment will also be required to complete the Safety Follow-up Visit, approximately 28 days after their last dose of study drug. The assessments performed at the Safety Follow-up Visit are listed in Table 3-2.

If the ETT Visit occurs 3 weeks or later following the last dose of study drug, then the ETT Visit will replace the Safety Follow-up Visit, and a separate Safety Follow-up Visit will not be required.

If a subject withdraws from the study and also withdraws consent or assent, no further assessments will be performed. Vertex may retain and continue to use any data and samples collected before such withdrawal of consent or assent.

## 9.1.5.1 Discontinuation During the Run-in Period

Subjects who prematurely discontinue study drug treatment during the Run-in Period will not be randomized or participate in the Treatment Period. These subjects will complete an ETT Visit and Safety Follow-up Visit (as applicable; see Section 9.1.5). The Safety Follow-up Visit will be their last visit in the study.

## 9.1.5.2 Discontinuation During the Treatment Period

Subjects who prematurely discontinue study drug treatment during the Treatment Period will continue to complete all scheduled study visits for assessments following completion of the ETT Visit, as detailed in Table 3-2.

These subjects will

complete an ETT Visit and Safety Follow-up Visit (as applicable; see Section 9.1.5). The Safety Follow-up Visit will be their last visit in the study.

#### 9.1.6 Lost to Follow-up

A subject will be considered lost to follow-up if both of the following occur:

- The subject misses 2 consecutive study visits (telephone contact and/or clinic visit) and is subsequently unable to be contacted by telephone (3 documented attempts by telephone within 2 weeks following the second missed visit)
- The subject does not respond within 2 weeks to a registered letter sent after the 3 attempted telephone contacts.

## 9.1.7 Completion of Study Participation

Completion of study participation for each individual subject is defined as one of the following:

- For subjects who complete the Treatment Period and enter an open-label study within 28 days of the Week 4 Visit: the Week 4 Visit
- For subjects who complete the Treatment Period and do not enter an open-label study within 28 days of the Week 4 Visit: the Safety Follow-up Visit
- For subjects who prematurely discontinue study drug treatment during the Treatment Period but do not withdraw consent (and assent, as applicable): The ETT or Safety Follow-up Visit (if required)
- For subjects who prematurely discontinue study drug treatment during the TEZ/IVA Run-in Period but do not withdraw consent (and assent, as applicable): the ETT or Safety Follow-up Visit (if required)
- For subjects who withdraw consent or assent: date of withdrawal of consent or assent, whichever is earlier (Section 9.9)

If subjects are lost to follow-up (Section 9.1.6), the date of completion of study participation will be defined as the date of the last contact.

The end of study is defined in Section 13.2.8.

#### 9.1.8 Independent Data Monitoring Committee

This study will be monitored by an independent data monitoring committee (IDMC), which will conduct periodic reviews of safety data from the study (Section 12.3.6.2). Procedural details of the IDMC structure and function, frequency of meetings, and data planned for review will be included in the IDMC charter. The IDMC charter will be finalized before the first subject is screened.

## 9.2 Method of Assigning Subjects to Treatment Groups

Subjects will be randomized (1:1) to the TC VX-659/TEZ/IVA arm or to the TEZ/IVA arm. Randomization will be stratified by ppFEV<sub>1</sub> determined during the TEZ/IVA Run-in Period (Day -14 assessment; <70 versus  $\geq$ 70) and age at the Screening Visit (<18 versus  $\geq$ 18 years of age). If the Day -14 ppFEV<sub>1</sub> value is not valid or not available, the most recent available ppFEV<sub>1</sub> value will be used for stratification.

An interactive web response system (IWRS) will be used to assign subjects to treatment. The randomization code list will be produced by Vertex Biometrics or a qualified randomization vendor.

## 9.3 Rationale for Study Design and Study Drug Regimens

## 9.3.1 Study Design

This Phase 3 study will assess the efficacy, PD, safety, and PK of VX-659/TEZ/IVA TC therapy in subjects with CF who have an F/F genotype.

A randomized, double-blind, controlled study design was selected to ascertain the effects of VX-659/TEZ/IVA while avoiding observer bias. TEZ/IVA is considered an appropriate active control since the efficacy and safety of TEZ/IVA in F/F subjects have been demonstrated in Study VX14-661-106 (Study 661-106). Study 661-106 met its primary endpoint of absolute change in ppFEV<sub>1</sub> through Week 24, with a 4.0 percentage point treatment difference between TEZ/IVA and placebo. In Study 661-106, TEZ/IVA was well tolerated and no safety concerns attributable to TEZ/IVA were identified.

A 4-week TEZ/IVA Run-in Period was incorporated into this study to establish a reliable on-treatment (TEZ/IVA) baseline for comparison during the Treatment Period.

The study will have a 4-week treatment duration because previous studies of CFTR modulators (IVA, LUM/IVA, and TEZ/IVA) have demonstrated that efficacy related to lung function (ppFEV<sub>1</sub>) can be reliably established using an endpoint at Week 4. In these studies, rapid improvements in ppFEV<sub>1</sub> are observed by Day 15, with a separation between the active treatment and placebo groups that is sustained through 24 weeks of treatment. These studies were conducted in patients with different genotypes, baseline ppFEV<sub>1</sub>, and age groups, using CFTR modulators that had different magnitudes of response.

The extent of response to CFTR modulator treatment may depend on the subject's ppFEV<sub>1</sub> value (an index of disease severity) before the start of TC study drug dosing. Some subjects in this study may be receiving treatment with LUM/IVA or TEZ/IVA at Screening, while some subjects may not be receiving treatment with CFTR modulators. Therefore, randomization will be stratified by ppFEV<sub>1</sub> value determined during the TEZ/IVA Run-in Period after at least 13 days of TEZ/IVA (Day -14 assessment). Randomization will also be stratified by age at screening. This will ensure a balanced evaluation of adult and pediatric subjects.

## 9.3.2 Study Drug Dose

#### VX-659 Dosage

A VX-659 dose of 240 mg qd was selected for the current study based on an assessment of the benefit-risk profile from the ongoing Phase 2 Study VX16-659-101 (Study 659-101) Part 1,



#### **TEZ and IVA Dosages**

TEZ will be administered as 100 mg qd and IVA will be administered as 150 mg q12h. This is the approved dosing regimen for Symdeko, which is now approved in the US.

## 9.3.3 Rationale for Study Population

This study will enroll CF subjects with the F/F genotype. F/F patients have continuing unmet need despite the availability of CFTR modulators and are expected to respond to a TC regimen of VX-659/TEZ/IVA based on results from Phase 1 and 2 studies in subjects with a single responsive *F508del* allele (F/MF genotypes) and in vitro experiments in relevant human F/F cell-based model systems.

The VX-659 Phase 2 clinical safety and efficacy data support the enrollment of pediatric subjects ≥12 and <18 years of age in this study.

## 9.3.4 Rationale for Study Assessments

The PD and efficacy endpoints being evaluated (SwCl, spirometry, and patient-reported outcomes) are widely accepted and generally recognized as reliable, accurate, and relevant to the study of individuals with CF. SwCl was evaluated in the registration study of IVA (Kalydeco), and spirometry and CFQ-R assessments were evaluated in the registration studies of IVA (Kalydeco) and LUM/IVA combination therapy (Orkambi).





## 9.4 Study Restrictions

## 9.4.1 Prohibited Medications

Table 9-2 lists prohibited medications. A non-exhaustive list of study prohibitions and cautions for medication will be provided in the Study Reference Manual.

**Table 9-2** Prohibited Medications

| | Timing of Restriction | | |
|---|---|---|---|
| Medication | Start of Restriction | End of<br>Restriction | Rationale |
| Moderate and strong<br>CYP3A or CYP2C9<br>inducers | None allowed<br>within 14 days<br>before the first dose<br>of the study drug on<br>Day -28 | None allowed<br>through<br>completion of<br>study<br>participation | VX-659, TEZ, and IVA are metabolized extensively via CYP3A4. VX-659 is also metabolized by CYP2C9. Therefore, use of moderate and strong inducers of CYP3A or CYP2C9 and moderate and strong inhibitors of |
| Moderate and strong CYP3A inhibitors (except ciprofloxacin) <sup>a</sup> | None allowed<br>within 14 days<br>before the first dose<br>of the study drug on<br>Day -28 | None allowed<br>through<br>completion of<br>study<br>participation | CYP3A, which have the potential to alter the exposure of VX-659, TEZ, or IVA, will be prohibited. |
| Sensitive OATP1B1 substrates | None allowed<br>within 14 days<br>before the first dose<br>of the study drug on<br>Day -28 | None allowed<br>through<br>completion of<br>study<br>participation | VX-659 is a potential inhibitor of the hepatic transporter OATP1B1. Therefore, sensitive substrates of OATP1B1, such as HMG-CoA reductase inhibitors ("statins") are prohibited during treatment. |
| Non-Vertex CFTR<br>modulators<br>(investigational or<br>approved) | None allowed<br>within 28 days or<br>5 terminal half-lives<br>(whichever is<br>longer) before<br>screening | None allowed<br>through<br>completion of<br>study<br>participation | These agents may confound the results of this study. |
| Vertex CFTR<br>modulators<br>(investigational or<br>approved), except<br>for study drugs | None allowed from<br>the first dose of<br>study drug on<br>Day -28 | None allowed<br>until after the last<br>dose of study<br>drug | These agents may confound the results of this study. |

CYP: cytochrome P450; IVA: ivacaftor; OATP1B1: organic anion transporting polypeptide 1B1; TEZ: tezacaftor <sup>a</sup> Ciprofloxacin is not a moderate CYP3A inhibitor on the basis of results of a drug-drug interaction study conducted with IVA, a sensitive CYP3A substrate (Kalydeco [ivacaftor] US Package Insert).

#### 9.4.2 Exposure to Sunlight

Subjects will take appropriate measures to minimize exposure to UV radiation (e.g., prolonged sunlight, tanning booths) from Day 1 through completion of study participation.

#### 9.5 Prior and Concomitant Medications

Information regarding prior and concomitant medications, including CF medications, other medications, and herbal and naturopathic remedies, will be collected from each subject's source documentation for medications taken within 56 days before the Screening Visit through completion of study participation, as defined in Section 9.1.7.

For subjects who are screened but are not subsequently randomized into the Treatment Period, details of prior medication will be documented only in the subjects' source documents.

• Subjects should remain on a stable treatment regimen for their CF from 28 days before the TEZ/IVA Run-in/Day -28 through completion of study participation. Stable treatment regimen is defined as the current treatment regimen for CF that subjects have been following

for at least 28 days before the TEZ/IVA Run-in/Day -28. Subjects may remain on Vertex CFTR modulators (investigational or approved) during the Screening Period and may transition directly to the TEZ/IVA Run-in/Day -28 without a washout (Table 9-2). Subjects should not initiate long-term treatment with new medication from 28 days before the TEZ/IVA Run-in/Day -28 through completion of study participation. Guidelines for stable treatment regimens for CF are as follows:

- o Subjects who are taking inhaled tobramycin or other chronically inhaled antibiotics should remain on that regimen throughout the study.
- o Subjects who cycle onto and off of an inhaled antibiotic should continue on their prior schedule. The timing of the first dose of study drug on the Day 1 Visit should be synchronized as closely as possible (e.g., not more than  $\pm$  3 days) to the first day in the cycle onto the inhaled antibiotic.
- o Subjects who alternate between 2 different inhaled antibiotics should remain on the same cycling schedule during the study. The timing of the first dose of study drug on the Day 1 Visit should be synchronized as closely as possible (e.g., not more than ± 3 days) to the first day in the cycle onto 1 of the inhaled antibiotics.
- Subjects may receive doses of prednisone or prednisolone of up to 10 mg/day chronically, or up to 60 mg daily for up to 5 days.
- Information about bronchodilator use during the study will be collected and documented. Subjects who are using a bronchodilator must have their spirometry assessments performed according to the guidelines provided in Section 11.6.1.

## 9.6 Administration

#### **9.6.1** Dosing

Study drug will be administered orally. All subjects will receive the same number of tablets each day to maintain the blind. Additional information is provided in the Pharmacy Manual.

Study drug will be administered with a fat-containing meal or snack, such as a standard "CF" meal or snack or a standard meal.

- 1. It is recommended that the dose be taken within 30 minutes of the start of the meal or snack.
- 2. Study drug will be administered as fixed-dose combination (FDC) tablet(s) (e.g., 2 TC or matching placebo tablets; 1 TEZ/IVA or matching placebo tablet) in the morning and as 1 IVA tablet in the evening. For each subject, doses of study drugs will be taken at approximately the same time (± 2 hours) each day.
- 3. The date, amount taken, and time of study drug administration, including whether food was taken with each dose, will be recorded for the 2 doses before PK sample collection and the dose received on the morning of PK sample collection (if applicable).
- 4. On days of scheduled visits, the morning dose of study drug (TC, TEZ/IVA, or placebo) will be administered at the site after predose assessments have been completed. A meal or snack will be provided by the site for the morning dose of TC, TEZ/IVA, or placebo.
- 5. If a subject's scheduled visit is to occur in the afternoon, the following guidelines must be used:

- If the dose in the clinic will be within 6 hours of the subject's scheduled morning dose, the subject should withhold their morning dose of TC, TEZ/IVA, or placebo and the morning dose will be administered in the clinic.
- If the dose in the clinic will be more than 6 hours after the subject's scheduled morning dose, the subject should take the morning dose of TC, TEZ/IVA, or placebo at home.
- 6. Subjects will be instructed to bring all used and unused materials associated with the study drug to the site; study drug will be dispensed at each visit, as appropriate.

#### 9.6.2 Missed Doses

## 9.6.2.1 Morning Dose of Study Drug

If a subject misses the morning dose of study drug (TC, TEZ/IVA, or placebo) and recalls within 6 hours, the subject should take his/her dose with food. If more than 6 hours but fewer than 12 hours have elapsed after his/her usual dosing time, the subject should take the morning dose of TC, TEZ/IVA, or placebo but skip the evening dose of study drug (IVA). If more than 12 hours have elapsed after his/her usual dosing time, the subject should skip the morning dose of TC, TEZ/IVA, or placebo and take the evening dose of IVA.

## 9.6.2.2 Evening Dose of Study Drug

If a subject misses the evening dose of IVA and recalls within 6 hours, the subject should take his/her dose with food. If more than 6 hours have elapsed after his/her usual dosing time, the subject should skip that dose and resume his/her normal schedule for the following dose.

## 9.7 Dose Modification for Toxicity

No dose modifications for toxicity are allowed. Treatment may be interrupted as outlined in Section 9.8. If any unacceptable toxicity arises, individual subjects will discontinue dosing (Section 9.1.5).

## 9.8 Study Drug Interruption and Stopping Rules

The medical monitor should be notified of an interruption of study drug that lasts >72 hours for any reason and of the resumption of study drug after such interruption.

#### 9.8.1 Liver Function Tests

The central laboratory will notify the medical monitor of ALT or AST  $>3 \times$  ULN and total bilirubin  $>2 \times$  ULN that are derived from centrally submitted samples.

Subjects with new treatment-emergent ALT or AST elevations of  $>3 \times ULN$ , with or without total bilirubin  $>2 \times ULN$ , must be followed closely, including confirmatory testing performed by the central laboratory within 48 to 72 hours of the initial finding and subsequent close monitoring of ALT, AST, and bilirubin levels, as clinically indicated.

If a subject cannot return to the site for confirmatory testing, a local laboratory may be used. Local laboratory results must be reported immediately to the medical monitor, and the subject must have the tests repeated and sent to the central laboratory as soon as possible (ideally within 48 to 72 hours).

Study drug administration <u>must be interrupted</u> immediately (prior to confirmatory testing) if any of the following criteria are met:

- ALT or AST  $> 8 \times ULN$
- ALT or AST >5 × ULN for more than 2 weeks
- ALT or AST >3 × ULN, in association with total bilirubin >2 × ULN and/or clinical jaundice

A thorough investigation of potential causes should be conducted, and the subject should be followed closely for clinical progression.

Study drug administration **must be discontinued** if the following criterion is met:

• Subsequent ALT or AST values confirm the initial elevation that satisfied the interruption rule (above), and no convincing alternative etiology (e.g., acetaminophen use, viral hepatitis, alcohol ingestion) is identified, regardless of whether transaminase levels have improved

All subjects in whom treatment is discontinued for elevated transaminases (and bilirubin, as applicable) should have these levels monitored closely until levels normalize or return to baseline

If an alternative, reversible cause of transaminase elevation with or without increased bilirubin or clinical jaundice has been identified, study drug administration may be resumed once transaminases return to baseline or are  $\leq 2 \times ULN$ , whichever is higher. Regardless of the duration of interruption, the medical monitor should be notified prior to resumption of study drug. Upon resumption of study drug, transaminases and bilirubin should be assessed weekly for 4 weeks. If a protocol-defined transaminase elevation interruption threshold recurs within 4 weeks of rechallenge with the study drug (with confirmation of the initial elevation by repeat testing within 48 to 72 hours), then the study drug must be permanently discontinued, regardless of the presumed etiology.

#### 9.8.2 Rash

Individuals who develop a generalized rash will be monitored closely. Study drug dosing should be interrupted if a subject develops a generalized rash of Grade 3 or higher, or a rash that is considered a serious adverse event. The investigator will notify the medical monitor of any rash that results in interruption of study drug, is Grade 3 or higher (Section 13.1.1.4), or is a serious adverse event (SAE). Investigators should consider additional evaluation including laboratory testing (e.g., complete blood count [CBC] with differential, LFTs), photographs of the rash, and dermatology consultation. The investigator may consider resumption of study drug if considered clinically appropriate.

#### 9.9 Removal of Subjects

Subjects may withdraw from the study at any time at their own request. Subjects may be withdrawn from study drug treatment at any time at the discretion of the investigator or Vertex for safety, behavior, noncompliance with study procedures, or administrative reasons. If a subject

has been withdrawn from study drug treatment, the subject will continue to be followed, provided that the subject has not withdrawn consent (and assent, as applicable).

In addition, a subject must be discontinued from study drug treatment if the subject meets any of the following criteria:

- Has a screening *CFTR* genotype that does not confirm study eligibility if a previous *CFTR* genotype laboratory report was used to establish eligibility. These subjects must be discontinued from the study (Section 8.1)
- Meets any of the stopping (discontinuation) criteria (Section 9.7)
- Becomes pregnant (Section 11.7.7.2)

Subjects who discontinue study drug treatment should return for study assessments, as noted in Section 9.1.5.2.

If a subject does not return for a scheduled visit, reasonable effort will be made to contact the subject. In any circumstance, reasonable effort will be made to document subject outcome. The investigator will inquire about the reason for withdrawal, request that the subject return all unused investigational product(s), request that the subject return for an ETT Visit and Safety Follow-up Visit, if applicable (see Section 9.1.5), and follow up with the subject regarding any unresolved AEs.

If the subject withdraws consent or assent for the study, no further assessments will be performed. Vertex may retain and continue using the study data and samples after the study is over, and may use the samples and information in the development of the study compound, and for other drugs and diagnostics, in publications and presentations, and for education purposes. If the subject withdraws from the study, the study data and samples collected will remain part of the study. A subject will not be able to request the withdrawal of his/her information from the study data. A subject may request destruction of the samples collected from him/her during the study as long as those samples can be identified as his/her samples.

#### 9.10 Replacement of Subjects

Subjects who withdraw or are withdrawn before the first dose of study drug on Day 1 of the Treatment Period may be replaced.

Subjects who withdraw or are withdrawn for nonsafety reasons during the study drug treatment period(s) may be replaced at Vertex's discretion.

#### 10 STUDY DRUG INFORMATION AND MANAGEMENT

During the TEZ/IVA Run-in Period, study drug refers to TEZ/IVA and IVA.

During the Treatment Period, study drug refers to VX-659/TEZ/IVA and matching placebo, TEZ/IVA and matching placebo, and IVA.

#### 10.1 Preparation and Dispensing

Study drug may be dispensed only under the supervision of the investigator or an authorized designee and only for administration to the study subjects.

## 10.2 Packaging and Labeling

Study drug tablets will be supplied in blister cards by Vertex. Study drug labeling will be in compliance with applicable local and national regulations. Additional details regarding packaging, labeling, and dispensing for study drug will be in the Pharmacy Manual.

#### 10.3 Study Drug Supply, Storage, and Handling

VX-659/TEZ/IVA will be supplied as 2 FDC film-coated tablets (120 mg VX-659/50 mg TEZ/75 mg IVA). Matching VX-659/TEZ/IVA placebo tablets will be of similar size and appearance and contain 0-mg VX-659, 0-mg TEZ, and 0-mg IVA (Table 10-1).

TEZ/IVA will be supplied as an FDC film-coated tablet (100 mg TEZ/150 mg IVA). A matching TEZ/IVA placebo tablet will be of similar size and appearance and contain 0-mg TEZ and 0-mg IVA (Table 10-1).

IVA (150 mg) will be supplied as a tablet containing 150-mg IVA.

Blister cards must be stored under conditions noted in the Pharmacy Manual. The investigator, or an authorized designee (e.g., a licensed pharmacist), will ensure that all investigational product is stored in a secured area, under recommended storage conditions, and in accordance with applicable regulatory requirements. To ensure adequate records, all study drugs will be accounted for via the drug accountability forms as instructed by Vertex.

Table 10-1 Study Drug: Strength/Dosing Form/Route

| Drug Name, Dosing Form, Route | Strength |
|-----------------------------------------------|----------|
| VX-659/TEZ/IVA, FDC tablet, oral | |
| VX-659 | 120 mg |
| TEZ | 50 mg |
| 13.7 Å | 75 |
| IVA | 75 mg |
| VX-659/TEZ/IVA-matching placebo, tablet, oral | 0 mg |
| TEZ/IVA, FDC tablet, oral | |
| TEZ | 100 mg |
| IVA | 150 mg |
| TEZ/IVA-matching placebo, tablet, oral | 0 mg |
| IVA, tablet, oral | 150 mg |

FDC: fixed-dose combination; IVA: ivacaftor; TEZ: tezacaftor

## 10.4 Drug Accountability

The pharmacist or designated study site staff will maintain information regarding the dates and amounts of (1) study drug received; (2) study drug dispensed to the subjects; and (3) study drug returned by the subjects. Subjects will be instructed to return all used and unused materials associated with the study drug to the site. These materials will be retained at the site according to instructions provided by Vertex or its designee. The study monitor will review study drug records and inventory throughout the study.

If a site uses a site-specific drug accountability system and/or process, including processes associated with the destruction of returned materials, the process must be documented and

approved by Vertex. The study monitor must review the drug accountability documentation on a regular basis. The study monitor will promptly communicate to Vertex any discrepancies he/she is unable to resolve with the site.

## 10.5 Disposal, Return, or Retention of Unused Drug

The study site staff or pharmacy personnel will retain all materials returned by the subjects until the study monitor has performed drug accountability. The investigator will ensure that the materials are destroyed in compliance with applicable environmental regulations, institutional policy, and any special instructions provided by Vertex. Destruction will be adequately documented.

## 10.6 Compliance

To ensure treatment compliance, the investigator or designee will supervise all study drug dosing that occurs at the site. At each visit, site personnel will review that the subject is compliant with study drug dosing and remind the subject of study drug dosing requirements. Compliance will also be assessed by ongoing study drug count.

If a subject demonstrates continued noncompliance of study drug dosing despite educational efforts, the investigator should consider discontinuing the subject from the study.

## 10.7 Blinding and Unblinding

This will be a double-blind study.

## 10.7.1 Blinding

All subjects (and their parents/caregivers/companions), site personnel (including the investigator, the site monitor, and the study team), and members of the Vertex study team will be blinded to the treatment codes.

Individuals who may be unblinded include only the following:

- Any site personnel for whom this information is important to ensure the safety of the subject in the event of a life-threatening medical emergency
- Any site personnel for whom this information is important to ensure the safety of the subject and her fetus in the event of a pregnancy
- Vertex Global Patient Safety (GPS) and Regulatory Affairs personnel to satisfy SAE processing and reporting regulations
- Vendor preparing the final (production) randomization list
- Vertex IWRS Manager
- Vertex Clinical Supply Chain
- IDMC
- Vendor preparing the unblinded analysis of safety data for review by the IDMC
- Bioanalytical contract research organization (CRO) analyzing PK samples and the Vertex Bioanalytical personnel who is not a member of the study team but reviews raw data from the Bioanalytical CRO. The Vertex Bioanalytical study team member will continue to be blinded.
#### Access to Spirometry and SwCl Results:

During the conduct of the study, the Vertex study team will not have access to the spirometry or SwCl results after the first dose of study drug in the Treatment Period.

Shortly before any planned efficacy analysis is conducted, the spirometry and SwCl data will be reviewed for data cleaning purposes by a biostatistician who does not have access to the treatment codes.

Individual SwCl test results will not be disclosed to the study sites with the exception of the screening values. Subjects and their parents/caregivers/companions should not be informed of study-related spirometry results until Vertex has determined that the study has completed (i.e., CSR finalization), regardless of whether the subject has prematurely discontinued treatment.

## 10.7.2 Unblinding

At the initiation of the study, the study site will be instructed on the method for breaking the blind. The unblinding method will be either a manual or electronic process.

# **Unblinding of Individual Subject Treatment Assignments by Investigator for Medical Emergencies or Urgent Clinical Situations**

Unblinding of the individual subject's treatment by the investigator will be limited to medical emergencies or urgent clinical situations in which knowledge of the subject's study treatment is necessary for clinical management. In such cases, investigators will use their best judgment as to whether to unblind without first attempting to contact the medical monitor to discuss and agree to the need for unblinding. If investigators deem it not necessary to unblind immediately, they will first attempt to contact the medical monitor to discuss and agree to the need for unblinding. If investigators have tried but are unable to reach the medical monitor, they will use their best judgment, based on the nature and urgency of the clinical situation, and may proceed with unblinding without having successfully reached and discussed the situation with the medical monitor. In case of emergency, the investigator will have the final decision and unilateral right for unblinding.

Contact information for the medical monitor (or appropriate backup) will be provided in a separate document.

In addition, the Vertex Medical Information Call Center ( ) will answer calls 24 hours a day, 7 days a week, 365 days of the year, and will triage these calls to the study medical monitor or appropriate backup.

If a subject's treatment assignment has been unblinded for a medical emergency or urgent clinical situation, the medical monitor will be notified within 24 hours of the unblinding event. The reason and the date of the unblinding will be documented clearly in the subject's study file. Information about the treatment assignment obtained from the unblinding will be maintained in a secure location with controlled access and will not be shared with the sponsor (Vertex), CRO, or any site personnel (other than the physician treating the subject). In addition, the investigator will consider whether the clinical event that prompted unblinding will be considered an SAE, according to the regulatory definitions or criteria for SAEs, and if so, submit an SAE report to Vertex GPS or designee, per Section 13.1.2.

## Unblinding of Individual Subject Treatment Assignments by Vertex GPS or Designee for SAEs or Safety Concerns

Vertex GPS or designee will also unblind any SAE reports in compliance with regulatory reporting requirements. In addition, Vertex may, for matters relating to safety concerns, unblind individual subjects at any time.

#### 11 ASSESSMENTS

#### 11.1 Timing of Assessments

The timing of assessments is shown in Table 3-1 and Table 3-2.

## 11.2 Subject and Disease Characteristics

Subject and disease characteristics include the following: demographics, medical history, height, and weight.

Medical history will be elicited from each subject and extracted from medical records during screening. Based on the medical history, the subject will be assessed for any disqualifying medical conditions as specified in the inclusion and exclusion criteria. The medical history will include a complete review of systems, medical and surgical histories, and any allergies.

Height and weight will be measured with shoes off. Following screening, height will be collected only for subjects  $\leq 21$  years of age on the date of informed consent.

#### 11.3 Pharmacokinetics

## 11.3.1 Blood Sampling

Blood samples will be collected to determine plasma concentrations of VX-659, TEZ, M1-TEZ, and IVA.

The Day 1 predose PK sample must be collected before dosing. The Week 4 predose PK sample must be collected within 60 minutes before dosing for subjects who are receiving their first dose of study drug in an open-label study on the same day as the Week 4 Visit. For subjects who are not entering an open-label study on the same day as the Week 4 Visit, the Week 4 sample should be collected approximately 12 hours after the evening dose of IVA before the Week 4 Visit.

All efforts should be made to obtain the PK samples during this specified window. Samples collected outside of the window will be considered protocol deviations.

For each visit with a PK blood draw, a record of study drug administration will be collected as described in Section 9.6. The collection date and exact time that each PK blood sample is drawn will also be recorded.

Samples from the PK sampling will be kept frozen by Vertex or its designee until all analyses have been completed and then disposed of according to Vertex or designee standard operating procedures.

Plasma concentration samples collected from subjects treated with placebo will not be routinely analyzed.

## 11.3.2 Processing and Handling of Pharmacokinetic Samples

Detailed procedures for the collection of blood samples and further procedures for processing and handling of samples for PK analysis will be provided in the PK Sample Handling Guidelines.

## 11.3.3 Bioanalysis

Samples will be analyzed using validated analytical methods in compliance with Vertex or designee standard operating procedures. A description of the assays and validation data will be provided in separate reports.

### 11.4 Pharmacodynamics: Sweat Chloride

SwCl samples will be collected with an approved collection device. Each collection will occur before study drug dosing (Section 9.6.1). At each time point, 2 samples will be collected, 1 from each arm (left and right). Sweat samples will be sent to a central laboratory for testing and interpretation of results. Specific instructions for the collection, handling, processing, and shipping of SwCl samples to the central laboratory will be provided separately.

See Section 10.7.1 for information about access to SwCl results.





## 11.6 Efficacy

## 11.6.1 Spirometry

Spirometry will be performed according to the American Thoracic Society Guidelines/European Respiratory Society Guidelines<sup>10</sup> and according to the additional guidelines that follow.

Pre-bronchodilator spirometry is defined as spirometry testing performed for subjects who have

- withheld their short-acting bronchodilators (e.g., albuterol) or anticholinergic (e.g., ipratropium bromide [Atrovent®]) for more than 4 hours before the spirometry assessment;
- withheld their long-acting bronchodilator (e.g., salmeterol) for more than 12 hours before the spirometry assessment; and
- withheld their once-daily, long-acting bronchodilator (e.g., tiotropium bromide [Spiriva®]) for more than 24 hours before the spirometry assessment.

During the Screening Period, spirometry assessments may be performed pre- or post-bronchodilator. At all other visits, all spirometry assessments should be performed pre-bronchodilator. During the Treatment Period, spirometry assessments must be performed before study drug dosing (Section 9.6.1) at approximately the same time at each visit. In the

event that a subject forgets to withhold bronchodilator(s), spirometry should be performed according to the following:

- If a subject's Day 1 spirometry assessment is pre-bronchodilator, but, on a subsequent visit, the subject forgets to withhold bronchodilator use, a post-bronchodilator spirometry assessment will be obtained for that visit only, and the visit will not be rescheduled.
- If, on Day 1, the subject forgets to withhold his/her dose of bronchodilator, spirometry should be performed post-bronchodilator, and all subsequent spirometric measurements (according to the schedule of assessments in Table 3-2) should be performed post-bronchodilator.
- Each spirometry assessment will be recorded in the source documents as pre- or post-bronchodilator.

All sites will be provided with spirometers to be used for all study assessments. Spirometry data will be transmitted to a centralized spirometry service for quality review. The investigator's assessment of the spirometry results will be used for the screening assessment and determination of eligibility.

See Section 10.7.1 for information about access to spirometry results.

The measured spirometric values listed below will be converted to percent predicted values using the standard equations of GLI.<sup>9</sup>

• FEV<sub>1</sub> (L)



#### 11.6.2 Cystic Fibrosis Questionnaire-Revised

The questionnaires provide information about demographics; general quality of life, school, work, or daily activities; and symptom difficulties (pertaining to CF).

Subjects will be asked to complete the CFQ-R in their native language, if validated translations are available. <sup>18, 19</sup> If there is no validated translation available in the subject's native language, the subject will not complete the questionnaire. Copies of the CFQ-R used will be provided in the Study Reference Manual. Validated translations of the CFQ-R, if available, will be provided for participating centers in non-English-speaking countries. <sup>20, 21</sup>

The CFQ-R will be completed before any other assessments are performed at that visit.

Subjects who are 12 and 13 years of age at the date of informed consent will complete the CFQ-R Child version themselves, and their parents/caregivers will complete the CFQ-R Parent version, at all visits, regardless of whether the subject subsequently turns 14 years of age during the study. Subjects 14 years of age and older at the date of informed consent will complete the Adolescent/Adult version of the questionnaire themselves at all visits.

#### 11.7 Safety

Safety evaluations will include AEs, clinical laboratory assessments, and clinical evaluation of vital signs, ECGs, PEs, and pulse oximetry.

For subjects <18 years of age on the date of informed consent, ophthalmological examinations will also be performed at screening (if not done within preceding 3 months).

#### 11.7.1 Adverse Events

All AEs will be assessed, documented, and reported in accordance with ICH GCP guidelines. Section 13.1 outlines the definitions, collection periods, criteria, and procedures for documenting, grading, and reporting AEs. A separate document that details AE case report form (CRF) completion guidelines for investigators as well as training will be provided.

#### 11.7.2 Clinical Laboratory Assessments

Blood and urine samples will be analyzed at a central laboratory, with the exception of the urine pregnancy tests. On Day -28 and Day 1, blood samples will be collected before the first dose of the study drug in the study period.

Laboratory test results that are abnormal and considered clinically significant will be reported as AEs.

The safety laboratory test panels are shown in Table 11-1.

**Table 11-1** Safety Laboratory Test Panels

| Serum Chemistry | Hematology | Urinalysis <sup>a</sup> |
|---|---|---|
| Glucose | Hemoglobin | Leukocyte esterase |
| Blood urea nitrogen <sup>b</sup> | Erythrocytes | Nitrite |
| Creatinine | Mean corpuscular volume | Urobilinogen |
| Sodium | Platelets | Urine protein |
| Potassium | Reticulocytes | pН |
| Calcium | Leukocytes | Urine blood |
| Chloride | Differential (absolute and percent): | Specific gravity |
| Magnesium | Eosinophils | Urine ketones |
| Bicarbonate | Basophils | Urine bilirubin |
| Inorganic phosphate | Neutrophils | Urine glucose |
| Total and direct bilirubin | Lymphocytes | |
| Alkaline phosphatase | Monocytes | |
| Aspartate transaminase | <b>Coagulation Studies</b> | |
| Alanine transaminase | Activated partial thromboplastin time | _ |
| Amylase | Prothrombin time | |
| Lipase | Prothrombin time International | |
| Gamma-glutamyl transferase | Normalized Ratio | |
| Protein | | |
| Albumin | | |
| Creatine kinase | | |
| Total cholesterol | | |
| Lactate dehydrogenase | | |

Note: Haptoglobin may be analyzed if judged to be clinically appropriate by the investigator.

Pregnancy (β-human chorionic gonadotropin) Tests for Females of Childbearing Potential: Any

If urinalysis results are positive for leukocyte esterase, nitrite, protein, or blood, microscopic examination of urine will be performed, and results will be provided for leukocytes, erythrocytes, crystals, bacteria, and casts.

If blood urea nitrogen cannot be collected, urea may be substituted.

female subject who does not meet the criteria for non-childbearing potential is considered to be of childbearing potential and must have a serum pregnancy test at screening. A definition of non-childbearing potential is provided in Section 11.7.7.1. Serum pregnancy tests will be performed at the study site and analyzed at the central laboratory. Urine pregnancy tests will be performed and analyzed at the site. The urine pregnancy test on Day -28 and Day 1 must be negative before the first dose of study drug in the study period. Additional pregnancy tests may be required according to local regulations and/or requirements.

<u>FSH (Screening Period Only)</u>: Blood samples for FSH will be measured for any suspected postmenopausal female with at least 12 months of continuous spontaneous amenorrhea. Serum FSH levels must be in the postmenopausal range as determined by the laboratory performing the test.

<u>CFTR Genotype (Screening Period Only):</u> CFTR genotyping will be performed for all subjects. If the screening CFTR genotype result is not received before Day -28, a previous CFTR genotype laboratory report may be used to establish eligibility. Subjects who have been enrolled and whose screening genotype is not confirmed to be F/F must be discontinued from the study (Section 9.9).

G6PD Activity Test (Screening Period Only): A blood sample will be collected for a quantitative G6PD activity assay, which will be performed in an established laboratory that runs the assay routinely. The use of a local laboratory that routinely runs the assay is permissible following approval by the medical monitor. In the event of a low G6PD activity result, the site will notify the Medical Monitor.

<u>Additional Evaluations</u>: Additional clinical laboratory evaluations will be performed at other times if judged to be clinically appropriate.

For the purposes of study conduct and unless noted otherwise (e.g., G6PD activity test), only laboratory tests done in the central laboratory may be used. Local laboratories may be used at the discretion of the local investigator for management of urgent medical issues. If a local laboratory test value is found to be abnormal and clinically significant, it will be verified by the central laboratory as soon as possible after the investigator becomes aware of the abnormal result. If it is not possible to send a timely specimen to the central laboratory (e.g., the subject was hospitalized elsewhere), the investigator may base the assessment of an AE on the local laboratory value.

## 11.7.3 Physical Examinations and Vital Signs

A PE of all body systems and vital signs assessment will be performed at screening and select study visits (see Table 3-1 and Table 3-2). At other visits, symptom-directed PEs and symptom-directed vital sign assessments will occur at any time if deemed necessary by the investigator or healthcare provider.

A complete PE includes a review of the following systems: head, neck, and thyroid; eyes, ears, nose, and throat (EENT); respiratory; cardiovascular; lymph nodes; abdomen; skin; musculoskeletal; and neurological. Breast, anorectal, and genital examinations will be performed when medically indicated. After screening, any clinically significant abnormal findings in PEs will be reported as AEs.

The abbreviated PE will include an assessment of the following body systems: EENT, cardiovascular system, respiratory system, skin, and abdomen.

Vital signs include blood pressure (systolic and diastolic), temperature (oral), pulse rate, and respiration rate. These will be assessed before dosing and following at least a 5-minute rest.

## 11.7.4 Pulse Oximetry

Pulse oximetry is a noninvasive measure of oxygen delivery to the tissues and has been correlated with clinical status and lung function. Arterial oxygen saturation by pulse oximetry will be assessed following at least a 5-minute rest and before study drug dosing. At visits when study drug is taken at the site, pulse oximetry will be collected before study drug dosing (Section 9.6.1).

## 11.7.5 Electrocardiograms

Standard 12-lead ECGs will be performed using a machine with printout according to the Schedule of Assessments (Table 3-1 and Table 3-2). Additional standard 12-lead ECGs will be performed at any other time if clinically indicated. Subjects will be instructed to rest for at least 5 minutes before having an ECG performed.

The ECG traces will be manually read at the study site. A printout of the ECG traces will be made for safety review by the investigator and maintained with source documentation. Clinically significant ECG abnormalities occurring during the study through completion of study participation will be recorded as AEs.

To ensure the safety of the subjects, a qualified individual at the study site will make comparisons to baseline measurements. If the QTcF is increased by >60 msec from the baseline or an absolute QTcF value is  $\geq 500$  msec for any scheduled ECG, 2 additional ECGs will be performed approximately 2 to 4 minutes apart to confirm the original measurement. If either of the QTcF values from these repeated ECGs remains above the threshold value (>60 msec from baseline or  $\geq 500$  msec), a single ECG will be repeated at least hourly until QTcF values from 2 successive ECGs fall below the threshold value that triggered the repeat measurement. Further details pertaining to ECGs will be provided to sites in the ECG Manual.

## 11.7.6 Ophthalmologic Examination

Ophthalmologic examinations will be conducted at screening only for subjects who are <18 years of age on the date of informed consent. The examination does not need to be completed if there is documentation of bilateral lens removal for the subject.

All examinations will be conducted by a licensed ophthalmologist or optometrist and will include

- measurement of best-corrected distance visual acuity of each eye; and
- pharmacologically dilated examination of the lens with a slit lamp

The screening examination does not need to be conducted if there is documentation of an examination meeting the protocol requirements that was conducted within 3 months before the date of informed consent.

Any clinically significant abnormal findings will be reported as AEs.

For subjects who subsequently enroll in an open-label study, follow-up ophthalmologic examinations will be performed as per that study's protocol.

## 11.7.7 Contraception and Pregnancy

The effects of VX-659 monotherapy or in TC with TEZ and IVA on conception, pregnancy, and lactation in humans are not known. VX-659, TEZ, and IVA did not show genotoxic potential in a standard battery of in vitro (Ames test, chromosomal aberration, or micronucleus in cultured mammalian cells) and in vivo (rodent micronucleus) studies. Reproductive toxicology studies of VX-659, TEZ, and IVA have not shown teratogenicity in rats and rabbits.

#### 11.7.7.1 Contraception

#### Contraception requirement for a couple is waived for the following:

- True abstinence for the subject, when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception. True abstinence must be practiced from the Screening Visit through 90 days after the last dose of study drug.
- If the male is infertile (e.g., bilateral orchiectomy). If a male subject is assumed to have complete bilateral absence of the vas deferens, infertility must be documented before the first dose of study drug (e.g., examination of a semen specimen or by demonstration of the absence of the vas deferens by ultrasound).
- If the female is of non-childbearing potential. To be considered of non-childbearing potential, the female must meet at least 1 of the following criteria:
  - o Postmenopausal: Amenorrheic for at least 12 consecutive months and a serum FSH level within the laboratory's reference range for postmenopausal females
  - o Documented hysterectomy or bilateral oophorectomy/salpingo-oophorectomy

Note: All other females (including females with tubal ligations) will be considered to be of childbearing potential.

• Same-sex relationships

For subjects for whom the contraception requirement is not waived, study participation requires a commitment from the subject that at least 1 acceptable method of contraception is used as a couple. Methods of contraception must be in successful use from signing of consent (or assent, when applicable), approximately 28 days before the first dose of study drug on Day -28 (unless otherwise noted), and until 90 days following the last dose of study drug. Additional contraception requirements may need to be followed according to local regulations and/or requirements. Acceptable methods of contraception are listed in Table 11-2.

Nob

Yes

Nob

Male Subjects and Their Female Subjects and Female (Non-study) Their Male (Non-study) **Partners Partners** Vasectomy performed at least 6 months previously, Yes Yes with a documented negative postvasectomy semen analysis for sperm Bilateral tubal occlusion (e.g., ligation) performed at Yes Yes least 6 months previously Male or female condom with or without spermicide<sup>a</sup> Yes Yes Female barrier contraception (such as diaphragm, Yes Yes cervical cap, or sponge) with spermicide Continuous use of an intrauterine device for at least 90 days before the first dose of study drug

**Table 11-2** Acceptable Methods of Contraception

Yes

Yes

Yes

#### **Additional notes:**

Hormone-releasing

Non-hormone releasing

Hormonal contraceptives, if successfully used for at

least 60 days before the first dose of study drug

- Male subjects must not donate sperm during the period starting from the first dose of study drug until 90 days after the last dose of study drug.
- Female subjects should not nurse a child during the period starting from the first dose of study drug until 90 days after the last dose of study drug.
- For male subjects with a female partner of childbearing potential, the couple should not plan to become pregnant during the study or within 90 days after the last dose of study drug, with the exception of couples who plan to become pregnant by artificial insemination using sperm banked by the male subject before the first dose of study drug or sperm from another source.

## **11.7.7.2 Pregnancy**

Subjects will be counseled to inform the investigator of any pregnancy that occurs during study treatment and for 90 days after the last dose of study drug.

If a female subject becomes pregnant during study participation, study drug will be permanently discontinued immediately. The investigator will notify the medical monitor and Vertex GPS within 24 hours of the site's knowledge of the subject's (or partner's) pregnancy using the Pregnancy Information Collection Form. Male subjects with female partners who become pregnant during the study must use a male condom to avoid exposure of a potential embryo or fetus to study drug via the seminal fluid.

The subject or partner will be followed until the end of the pregnancy and the infant will be followed for 1 year after the birth, provided informed consent is obtained. A separate ICF will be provided to explain these follow-up activities. Pregnancy itself does not constitute an AE.

<sup>&</sup>lt;sup>a</sup> A female condom cannot be used with a male condom due to risk of tearing.

Hormone-releasing intrauterine devices and hormonal contraceptives are <u>not</u> considered an acceptable method in female study subjects due to potential induction of metabolism by VX-659; however, female subjects are not required to discontinue their use of hormone-releasing intrauterine devices or hormonal contraceptives.

#### 12 STATISTICAL AND ANALYTICAL PLANS

This section presents a summary of the planned analyses for this protocol. Statistical analysis details will be provided in the statistical analysis plan (SAP), and clinical pharmacologic analysis details will be provided in the clinical pharmacology analysis plan (CPAP), both of which will be finalized before the clinical data lock for the study and treatment unblinding.

### 12.1 Sample Size and Power

The primary efficacy endpoint is the absolute change in  $ppFEV_1$  from baseline at Week 4. The primary null hypothesis to be tested is that the mean absolute change in  $ppFEV_1$  from baseline at Week 4 is the same for the TC and TEZ/IVA treatment groups. The null hypothesis will be tested at a 2-sided significance level of 0.05.

Assuming a within-group SD of 7 percentage points and a 5% dropout rate at Week 4, a sample size of 50 subjects in each treatment group for a total of 100 subjects will have approximately 93% power to detect a difference of 5.0 percentage points for the mean absolute change in ppFEV<sub>1</sub> from baseline at Week 4 between the 2 treatment groups, based on a 2-sided 2-sample *t*-test at a significance level of 0.05 using the PASS software (Version 11.0).

## 12.2 Analysis Sets

The following analysis sets are defined: All Subjects Set, Full Analysis Set (FAS), and Safety Set. Additional analysis sets related to the Run-in Period will be defined in the SAP, as appropriate.

The **All Subjects Set** will include all subjects who were randomized or received at least 1 dose of study drug. This analysis set will be used for all individual subject data listings and disposition summary tables, unless otherwise specified.

The **FAS** will include all randomized subjects who carry the intended *CFTR* allele mutation and receive at least 1 dose of study drug in the Treatment Period. The FAS will be used to summarize subject demographics and baseline characteristics, and for all efficacy analyses in which subjects will be analyzed according to their randomized treatment group, unless otherwise specified.

The **Safety Set** will include all subjects who received at least 1 dose of study drug in the Treatment Period. The Safety Set will be used for all safety analyses in which subjects will be analyzed according to the treatment they received, unless otherwise specified.

#### 12.3 Statistical Analysis

#### 12.3.1 General Considerations

Continuous variables will be summarized using the following descriptive summary statistics: the number of subjects (n), mean, SD, median, minimum value (min), and maximum value (max). The precision of the measurement for each continuous variable will be specified in the SAP. Unless otherwise specified, min and max values will be reported with the same precision as the units of the raw data. The mean, median, and SD will be reported to 1 additional decimal place. Any values that require a transformation to standard units (metric or SI) will be converted with the appropriate precision.

**Categorical variables** will be summarized using counts and percentages. Percentages will be presented to 1 decimal place.

The **baseline value**, unless otherwise specified, will be defined as the most recent non-missing measurement (scheduled or unscheduled) collected before the first dose of study drug in the Treatment Period (i.e., the Day 1 Visit). For ECG, baseline will be defined as the most recent pretreatment measurement (or the average of triplicate measurements, if the most recent pretreatment measurement is obtained in triplicate) before the first dose of study drug in the Treatment Period (i.e., the Day 1 Visit).

**Absolute change** from baseline will be calculated as post-baseline value – baseline value.

The **Treatment-emergent (TE) Period for the Run-in Period** will be from the first dose of study drug in the Run-in Period to (1) the first dose of study drug in the Treatment Period for subjects who complete the Run-in Period and continue to the Treatment Period, or (2) 28 days after the last dose date of study drug in the Run-in Period for subjects who do not continue to the Treatment Period (e.g., subjects who do not meet the conditions to enter the Treatment Period).

The **TE Period for the Treatment Period** will include the time from the first dose date of study drug in the Treatment Period (TC or placebo + TEZ/IVA) to 28 days after the last dose of the study drug or to the completion of study participation date (as defined in Section 9.1.7), whichever occurs first.

#### 12.3.2 Background Characteristics

## 12.3.2.1 Subject Disposition

The number and percentage of subjects in each disposition category (e.g., randomized, included in the FAS, included in the Safety Set, completed Treatment Period, completed study, prematurely discontinued treatment or study with a breakdown of the reasons for discontinuation, and entered an open-label study) will be summarized overall and by treatment group.

An additional subject disposition summary related to the TEZ/IVA Run-in Period will be defined in the SAP, as appropriate.

## 12.3.2.2 Demographics and Baseline Characteristics

Demographic, medical history, and baseline characteristics will be summarized using descriptive summary statistics.

The following demographics and baseline characteristics will be summarized overall and by treatment group for the FAS, and will include (but are not limited to): sex, race, baseline age, baseline weight, baseline height, baseline BMI, baseline ppFEV<sub>1</sub>, and baseline SwCl.

Medical history will be summarized by MedDRA System Organ Class (SOC) and Preferred Term (PT) for the FAS.

No statistical tests will be performed to evaluate baseline imbalance between treatment groups.

#### 12.3.2.3 Prior and Concomitant Medications

Medications will be coded using the World Health Organization Drug-Dictionary and categorized as follows:

• **Prior medication**: any medication that was administered during the 56 days before the first dose of study drug in the Treatment Period

- Concomitant medication during the Run-in Period: medication continued or newly received during the TE Period for the Run-in Period
- Concomitant medication during the Treatment Period: medication continued or newly received during the TE Period for the Treatment Period
- **Post-treatment medication**: medication continued or newly received after:
  - o the TE Period for the Run-in Period if the subject did not receive study drug in the Treatment Period
  - o the TE Period for the Treatment Period for subjects who received study drug in the Treatment Period

A given medication may be classified as a prior medication, a concomitant medication, or a post-treatment medication; both prior and concomitant; both concomitant and post-treatment; or prior, concomitant, and post-treatment. If a medication has a missing or partially missing start/end date or time and if it cannot be determined whether it was taken before the first dose of study drug, concomitantly during the TE Period, or after the TE Period, it will be considered in all 3 categories of prior, concomitant, and post-treatment medication.

Prior medications and concomitant medications will be summarized descriptively by Preferred Name, overall, and by treatment group based on the FAS. Post-treatment medications will be provided separately in an individual subject data listing.

#### 12.3.2.4 Study Drug Exposure and Compliance

Study drug exposure and compliance will be summarized for the Treatment Period only.

Study drug exposure will be summarized overall and by treatment group, based on the Safety Set in terms of the duration of treatment a subject received (in days), defined as the last day – the first day of study drug plus 1, regardless of study drug interruption.

Study drug compliance will be summarized overall and by treatment group based on the FAS, and will be calculated as:  $100 \times [1- (total number of days of study drug interruption) / (duration of study drug exposure in days)]. A study drug interruption on a given day is defined as an interruption of any study drug on that day.$ 

In addition, percentage of tablets taken will also be summarized overall and by treatment group based on the FAS, and will be calculated as  $100 \times [(\text{total number of tablets dispensed for the Treatment Period}) - (total number of tablets returned for the Treatment Period)] / (total number of tablets planned to be taken per day × duration of study drug exposure in days for the Treatment Period).$ 

#### 12.3.2.5 Important Protocol Deviations

An important protocol deviation (IPD) is a deviation that may significantly affect the completeness, accuracy, or reliability of the study data or that may significantly affect a subject's rights, safety, or well-being. The rules for identifying an IPD will be described in the SAP.

All IPDs will be provided in an individual subject data listing and summarized, as appropriate.

## 12.3.3 Efficacy and Pharmacodynamic Analyses

The primary objective of the study is the evaluation of the efficacy of VX-659 in TC with TEZ and IVA. The analysis in this section will be based on the FAS, unless otherwise specified.

## 12.3.3.1 Analysis of Primary Variable

The primary efficacy variable is the absolute change in ppFEV<sub>1</sub> from baseline at Week 4. The analysis of this variable will be performed using a mixed-effects model for repeated measures (MMRM) with absolute change from baseline in ppFEV<sub>1</sub> at Day 15 and Week 4 as the dependent variable. The model will include treatment group, visit, and treatment-by-visit interaction as fixed effects, with continuous baseline ppFEV<sub>1</sub> and age at screening (<18 versus  $\ge18$  years of age) as covariates. The model will be estimated using restricted maximum likelihood. Denominator degrees of freedom for the F test for fixed effects will be estimated using the Kenward-Roger approximation. An unstructured covariance structure will be used to model the within-subject errors. If the model estimation does not converge, a compound symmetry covariance structure will be used instead. Conditional on the observed data and covariates, missing data will be assumed to be missing at random; consequently, no imputation of missing data will be performed.

The primary result obtained from the model will be the estimated treatment difference at Week 4. The adjusted mean with a 2-sided 95% CI and a 2-sided *P* value will be provided. Furthermore, the treatment difference at each post-baseline visit will also be provided, obtained from the model.

## 12.3.3.2 Analysis of Key Secondary Variables

The key secondary variables are:

- Absolute change in SwCl from baseline at Week 4: Analysis of this pharmacodynamics
  (PD) variable will be based on an MMRM model similar to the analysis of the primary
  efficacy variable. Data obtained from the Day 15 and Week 4 Visits will be included in the
  model.
- Absolute change in the CFQ-R respiratory domain score from baseline at Week 4: Analysis of this domain will be based on an MMRM model similar to the analysis of the primary efficacy variable. Data obtained from the Day 15 and Week 4 Visits will be included in the model.

Details will be provided in the SAP.



## 12.3.3.4 Multiplicity Adjustment

A hierarchical testing procedure will be used to control the overall type I error at an alpha of 0.05 for the primary endpoint and the key secondary endpoints tested. The key secondary endpoints of absolute change in SwCl from baseline at Week 4 and absolute change in CFQ-R respiratory domain score from baseline at Week 4 will only be tested at an alpha of 0.05 if the primary endpoint of absolute change in ppFEV<sub>1</sub> from baseline at Week 4 is statistically significant. The second key secondary endpoint will only be tested if the first key secondary endpoint is statistically significant. The testing order of the key secondary endpoints is as follows:

- 1. First key secondary endpoint: Absolute change in SwCl from baseline at Week 4
- 2. Second key secondary endpoint: Absolute change in CFQ-R respiratory domain score from baseline at Week 4

## 12.3.4 Safety Analysis

All safety analyses will be based on data from the TE Period for all subjects in the Safety Set.

The overall safety profile of study drug will be assessed based on the following safety and tolerability endpoints:

- Treatment-emergent adverse events (TEAEs)
- Clinical laboratory values (i.e., hematology, serum chemistry, coagulation, and urinalysis)
- ECGs
- Vital signs
- Pulse oximetry

All safety data from the TE Period will be summarized by treatment group and overall.

All safety data will be presented in individual subject data listings, including safety data from the Run-in Period.

#### 12.3.4.1 Adverse Events

For analysis purposes, AEs will be classified as pretreatment AEs, TEAEs during the Run-in Period, TEAEs during the Treatment Period, or post-treatment AEs, defined as follows:

- **Pretreatment AE**: any AE that occurred before the first dose date of study drug (TEZ/IVA) in the Run-in Period
- **TEAE during the Run-in Period**: any AE that worsened (either in severity or seriousness) or that was newly developed at or after the first dose date of study drug (TEZ/IVA) through the end of the TE Period for the Run-in Period
- **TEAE during the Treatment Period**: any AE that worsened (either in severity or seriousness) or that was newly developed at or after the first dose date of study drug (TC or placebo + TEZ/IVA) through the end of the TE Period for the Treatment Period
- **Post-treatment AE**: any AE that worsened (either in severity or seriousness) or that was newly developed after:

- o the TE Period for the Run-in Period if the subject did not receive treatment in the Treatment Period
- o the TE Period for the Treatment Period if the subject received treatment in the Treatment Period

For AEs with missing or partial start dates, if there is no clear evidence that the AEs started before or after study drug treatment, then the AEs will be classified as TEAEs corresponding to the Treatment Period. Unless otherwise specified, TEAE refers to TEAE during the Treatment Period

AE summary tables will be presented for TEAEs, overall and by treatment group, and will include the following:

- All TEAEs
- TEAEs by strongest relationship
- TEAEs by maximum severity
- TEAEs leading to treatment discontinuation
- TEAEs leading to treatment interruption
- Grade 3 and Grade 4 TEAEs
- Serious TEAEs
- TEAEs leading to death
- Frequently reported TEAEs

Summaries will be presented by MedDRA SOC and PT using frequency counts and percentages (i.e., number and percentage of subjects with an event). When summarizing the number and percentage of subjects with an event, subjects with multiple occurrences of the same AE or a continuing AE will be counted once, only the maximum severity level will be presented in the severity summaries, and the strongest relationship level in the relationship summaries. In addition, a listing containing individual subject level AE data for all deaths and other serious and significant AEs will be provided separately. All AEs, including pre- and post-treatment AEs, will be presented in individual subject data listings.

## 12.3.4.2 Clinical Laboratory Assessments

For the treatment-emergent laboratory measurements, the observed values and change from baseline values of the continuous hematology, serum chemistry, and coagulation results will be summarized in SI units by treatment group at each visit.

The number and percentage of subjects with at least 1 threshold analysis event during the TE Period will be summarized overall and by treatment group. The threshold analysis criterion shift from baseline will also be summarized for select laboratory parameters. The threshold analysis criteria and the parameter selection criteria will be provided in the SAP.

Results of urinalysis and pregnancy tests will be listed in individual subject data listings only. In addition, a listing containing individual subject hematology, chemistry, and coagulation values outside the reference ranges will be provided. This listing will include data from scheduled and unscheduled visits.

## 12.3.4.3 Electrocardiogram

For the treatment-emergent ECG measurements, a summary of observed values and change from baseline values will be provided by treatment group, at each visit, as applicable, for the following ECG interval measurements (in msec): RR, PR, QT, and QT corrected for HR (QTcF), QRS duration, and HR (beats per minute).

The number and percentage of subjects with at least 1 threshold analysis event during the TE Period will be summarized overall and by treatment group. The threshold analysis criteria will be provided in the SAP.

Additional ECG analyses may be described in the SAP.

#### **12.3.4.4 Vital Signs**

For the treatment-emergent vital signs measurements, the observed values and change from baseline values will be summarized by treatment group at each visit. The following vital signs parameters will be summarized: systolic and diastolic blood pressure (mm Hg), body temperature (°C), pulse rate (beats per minute), and respiratory rate (breaths per minute).

The number and percentage of subjects with at least 1 threshold analysis event during the TE Period will be summarized overall and by treatment group. The threshold analysis criteria will be provided in the SAP.

Additional vital signs analyses may be described in the SAP.

#### 12.3.4.5 Pulse Oximetry

For the treatment-emergent pulse oximetry measurements, a summary of observed values and change from baseline values will be provided by treatment group, at each scheduled visit for the percent of oxygen saturation by pulse oximetry.

The number and percentage of subjects with shift changes from baseline (normal/missing and low according to the reference range) to the lowest percent of oxygen saturation during the TE Period will be summarized overall and by treatment group.

## 12.3.4.6 Physical Examination

PE findings will be presented in an individual subject data listing only.

## 12.3.4.7 Other Safety Analysis

Not applicable.



#### 12.3.6 Interim and IDMC Analyses

#### 12.3.6.1 Interim Analysis

Not applicable.

### 12.3.6.2 IDMC Analysis

The IDMC (Section 9.1.8) will conduct safety review of study data. Details will be described in the IDMC charter.

## 12.4 Clinical Pharmacology Analysis

#### 12.4.1 Pharmacokinetic Analysis

PK analysis of VX-659, TEZ, M1-TEZ, and IVA may be performed using nonlinear mixed-effects modeling, as data allow. Descriptive statistics will be used to summarize predose plasma concentrations for all analytes.

A detailed description of the planned PK analysis will be presented in the CPAP.

## 13 PROCEDURAL, ETHICAL, REGULATORY, AND ADMINISTRATIVE CONSIDERATIONS

# 13.1 Adverse Event and Serious Adverse Event Documentation, Severity Grading, and Reporting

#### 13.1.1 Adverse Events

#### 13.1.1.1 Definition of an Adverse Event

An AE is defined as any untoward medical occurrence in a subject during the study; the event does not necessarily have a causal relationship with the treatment. This includes any newly occurring event or worsening of a pre-existing condition (e.g., increase in its severity or frequency) after the ICF is signed.

An AE is considered serious if it meets the definition in Section 13.1.2.1.

#### 13.1.1.2 Clinically Significant Assessments

Study assessments including laboratory tests, ECGs, PEs, and vital signs will be assessed and those deemed to have clinically-significant worsening from baseline will be documented as an AE. When possible, a clinical diagnosis for the study assessment will be provided, rather than the abnormal test result alone (e.g., urinary tract infection, anemia). In the absence of a diagnosis, the abnormal study assessment itself will be listed as the AE (e.g., bacteria in urine or decreased hemoglobin).

An abnormal study assessment is considered clinically significant if the subject has 1 or more of the following:

- Concomitant signs or symptoms related to the abnormal study assessment
- Further diagnostic testing or medical/surgical intervention
- A change in the dose of study drug or discontinuation from the study

Repeat testing to determine whether the result is abnormal, in the absence of any of the above criteria, does not necessarily meet clinically significant criteria. The determination of whether the study assessment results are clinically significant will be made by the investigator.

A laboratory value that is Grade 4 will not automatically be an SAE. A Grade 4 laboratory value will be an SAE if the subject's clinical status indicates a life-threatening AE.

#### 13.1.1.3 Documentation of Adverse Events

All AEs will be collected from the time the ICF is signed until the subject completes study participation, as defined in Section 9.1.7.

All subjects will be queried, using nonleading questions, about the occurrence of AEs at each study visit. When possible, a constellation of signs and/or symptoms will be identified as 1 overall event or diagnosis. All AEs for enrolled subjects will be recorded in the CRF and source document. AEs for subjects who are screened but not subsequently enrolled in the study will be recorded only in the subject's source documents. The following data will be documented for each AE:

- Description of the event
- Classification of "serious" or "nonserious"
- Date of first occurrence and date of resolution (if applicable)
- Severity
- Causal relationship to study drug(s)
- Action taken
- Outcome
- Concomitant medication or other treatment given

## 13.1.1.4 Adverse Event Severity

The investigator will determine and record the severity of all serious and nonserious AEs. The guidance available at the following website will be consulted: Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0, Cancer Therapy Evaluation Program, http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm (Accessed 28 September 2017). AEs of CTCAE Grades 4 and 5 will be documented as "life-threatening." In considering the severity of an AE in a pediatric subject, the investigator will consider that reference ranges for pediatric clinical laboratory parameters may differ from those given in the CTCAE. The severity of an AE that does not appear in the CTCAE will be determined according to the definitions in Table 13-1.

Table 13-1 Grading of AE Severity

| Classification | Definition |
|---|---|
| Mild (Grade 1) | Mild level of discomfort and does not interfere with regular activities |
| Moderate (Grade 2) | Moderate level of discomfort and significantly interferes with regular activities |
| Severe (Grade 3) | Significant level of discomfort and prevents regular activities |
| Life-threatening (Grade 4) | Any adverse drug event that places the subject, in the view of the investigator, at immediate risk of death |

## 13.1.1.5 Adverse Event Causality

Every effort will be made by the investigator to assess the relationship of the AE, if any, to the study drug(s). Causality will be classified using the categories presented in Table 13-2.

Table 13-2 Classifications for AE Causality

| Classification | Definition |
|---|---|
| Related | There is an association between the event and the administration of investigational study drug, a plausible mechanism for the event to be related to the investigational study drug and causes other than the investigational study drug have been ruled out, and/or the event reappeared on re-exposure to the investigational study drug. |
| Possibly related | There is an association between the event and the administration of the investigational study drug and there is a plausible mechanism for the event to be related to investigational study drug, but there may also be alternative etiology, such as characteristics of the subject's clinical status or underlying disease. |
| Unlikely related | The event is unlikely to be related to the investigational study drug and likely to be related to factors other than investigational study drug. |
| Not related | The event is related to an etiology other than the investigational study drug (the alternative etiology will be documented in the study subject's medical record). |

## 13.1.1.6 Study Drug Action Taken

The investigator will classify the study drug action taken with regard to the AE. The action taken will be classified according to the categories shown in Table 13-3.

Table 13-3 Classifications for Study Drug Action Taken With Regard to an AE

| Classification | Definition |
|---|---|
| Dose not changed | Study drug dose not changed in response to an AE |
| Dose reduced | Study drug dose reduced in response to an AE |
| Drug interrupted | g interrupted Study drug administration interrupted in response to an AE |
| Drug withdrawn | Study drug administration permanently discontinued in response to an AE |
| Not applicable | Action taken regarding study drug administration does not apply. |
| | "Not applicable" will be used in circumstances such as when the investigational |
| | treatment had been completed before the AE began and no opportunity to decide |
| | whether to continue, interrupt, or withdraw treatment is possible. |

#### 13.1.1.7 Adverse Event Outcome

An AE will be followed until the investigator has determined and provided the final outcome. The outcome will be classified according to the categories shown in Table 13-4.

 Classification
 Definition

 Recovered/resolved
 Resolution of an AE with no residual signs or symptoms

 Recovered/resolved with sequelae
 Resolution of an AE with residual signs or symptoms

 Not recovered/not resolved (continuing)
 Either incomplete improvement or no improvement of an AE, such that it remains ongoing

 Fatal
 Outcome of an AE is death. "Fatal" will be used when death is at least possibly related to the AE.

Outcome of an AE is not known (e.g., a subject lost to follow-up)

Table 13-4 Classifications for Outcome of an AE

#### 13.1.1.8 Treatment Given

Unknown

The investigator ensures adequate medical care is provided to subjects for any AEs, including clinically significant laboratory values related to study drug. In addition, the investigator will describe whether any treatment was given for the AE. "Yes" is used if any treatment was given in response to an AE, and may include treatments such as other medications, surgery, or physical therapy. "No" indicates the absence of any kind of treatment for an AE.

#### 13.1.2 Serious Adverse Events

#### 13.1.2.1 Definition of a Serious Adverse Event

An SAE is any AE that meets any of the following outcomes:

- Fatal (death, regardless of cause, that occurs during participation in the study or occurs after participation in the study and is suspected of being a delayed toxicity due to administration of the study drug)
- Life-threatening, such that the subject was at immediate risk of death from the reaction as it occurred
- Inpatient hospitalization or prolongation of hospitalization
- Persistent or significant disability/incapacity (disability is defined as a substantial disruption of a person's ability to conduct normal life functions)
- Congenital anomaly or birth defect
- Important medical event that, based upon appropriate medical judgment, may jeopardize the subject or may require medical or surgical intervention to prevent 1 of the outcomes listed above (e.g., an allergic bronchospasm requiring intensive treatment in an emergency room or at home)

If a subject has a hospitalization or procedure (e.g., surgery) for an event or condition that occurred before the subject signed the ICF, and the hospitalization or procedure was planned before the subject signed the ICF, the hospitalization or procedure will not be considered to indicate an SAE, unless an AE caused the hospitalization or procedure to be rescheduled sooner or to be prolonged relative to what was planned. In addition, hospitalizations clearly not associated with an AE (e.g., social hospitalization for purposes of respite care) will not be considered to indicate an SAE.

Clarification will be made between the terms "serious" and "severe" because they are not synonymous. The term "severe" is often used to describe the intensity (severity) of a specific event, as in mild, moderate, or severe myocardial infarction. The event itself, however, may be of relatively minor medical significance, such as a severe headache. This is not the same as "serious," which is based on subject/event outcome or action described above, and is usually associated with events that pose a threat to a subject's life or functioning. Seriousness, not severity, serves as a guide for defining expedited regulatory reporting obligations.

#### 13.1.2.2 Documentation of Serious Adverse Events

All SAEs that occur after obtaining informed consent through completion of study participation, regardless of causality, will be reported by the investigator to Vertex GPS. In addition, all SAEs that occur after completion of study participation and are considered related to study drug(s) will be reported to Vertex GPS within 24 hours.

SAEs will be recorded on the Vertex Organized Safety Information Collection Form (hereafter referred to as the "SAE Form") using a recognized medical term or diagnosis that accurately reflects the event. SAEs will be assessed by the investigator for relationship to the investigational study drug(s) and possible etiologies. On the SAE Form, relationship to study drug(s) will be assessed only as related (includes possibly related) or not related (includes unlikely related), and severity assessment will not be required. For the purposes of study analysis, if the event has not resolved at the end of the study reporting period, it will be documented as ongoing. For purposes of regulatory safety monitoring, the investigator is required to follow the event to resolution and report to Vertex the outcome of the event using the SAE Form.

## 13.1.2.3 Reporting Serious Adverse Events

The investigator is responsible for notifying the sponsor within 24 hours of identifying an SAE, regardless of the presumed relationship to the investigational study drug. The SAE Form will be completed for new/initial events as well as to report follow-up information on previously reported events. Investigators are asked to report follow-up information as soon as it becomes available to ensure timely reporting to health authorities.

Email: (preferred choice)

Fax: For questions, contact telephone:

Please send completed SAE Forms to Vertex GPS via:

## 13.1.2.4 Expedited Reporting and Investigator Safety Letters

Vertex, as study sponsor, is responsible for reporting suspected, unexpected, serious adverse reactions (SUSARs) involving the study drug(s) to all regulatory authorities, IECs, and participating investigators in accordance with ICH Guidelines and/or local regulatory requirements, as applicable. In addition, Vertex, or authorized designee, will be responsible for the submission of safety letters to central IECs.

It is the responsibility of the investigator or designee to promptly notify the local IRB/local IEC of all unexpected serious adverse drug reactions involving risk to human subjects.

## 13.2 Administrative Requirements

#### 13.2.1 Ethical Considerations

The study will be conducted in accordance with the current ICH GCP guidelines, which are consistent with the ethical principles founded in the Declaration of Helsinki, and in accordance with local applicable laws and regulations. The IRB/IEC will review all appropriate study documentation to safeguard the rights, safety, and well-being of the subjects. The study will only be conducted at sites where IRB/IEC approval has been obtained. The protocol, Investigator's Brochure, sample ICF, advertisements (if applicable), written information given to the subjects (including diary cards), safety updates, annual progress reports, and any revisions to these documents will be provided to the IRB/IEC by the investigator or Vertex, as allowable by local applicable laws and regulations.

## 13.2.2 Subject Information and Informed Consent

After the study has been fully explained, written informed consent will be obtained from the subject or legal representative or guardian (if applicable), and assent will be obtained from the subject (if applicable), before study participation. The method of obtaining and documenting the informed consent and assent (if applicable) and the contents of the consent will comply with ICH GCP and all applicable laws and regulations and will be subject to approval by Vertex or its designee. When determining the age of the subject, other study eligibility criteria, and timing of collection applicable assessments, the informed consent will be used as the reference (e.g., age at time of informed consent, date of informed consent, timing of AE collection).

## 13.2.3 Investigator Compliance

No modifications to the protocol will be made without the approval of both the investigator and Vertex. Changes that significantly affect the safety of the subjects, the scope of the investigation, or the scientific quality of the study (i.e., efficacy assessments) will require IRB/IEC notification before implementation, except where the modification is necessary to eliminate an apparent immediate hazard to human subjects. Vertex will submit all protocol modifications to the required regulatory authorities.

When circumstances require an immediate departure from procedures set forth in the protocol, the investigator will contact Vertex to discuss the planned course of action. If possible, contact will be made before the implementation of any changes. Any departures from the protocol will be fully documented in the source documentation and in a protocol deviation log.

#### 13.2.4 Access to Records

The investigator will make the office and/or hospital records of subjects enrolled in this study available for inspection by Vertex or its representative at the time of each monitoring visit and for audits. The records will also be available for direct inspection, verification, and copying, as required by applicable laws and regulations, by officials of the regulatory health authorities (FDA and others). The investigator will comply with applicable privacy and security laws for use and disclosure of information related to the research set forth in this protocol.

#### 13.2.5 Subject Privacy

To maintain subject confidentiality and to comply with applicable data protection and privacy laws and regulations, all CRFs, study reports, and communications relating to the study will identify subjects by assigned subject numbers and access to subject names linked to such

numbers shall be limited to the site and the study physician and shall not be disclosed to Vertex. As required by applicable laws and regulations in the countries in which the study is being conducted, the investigator will allow Vertex and/or its representatives access to all pertinent medical records to allow for the verification of data gathered in the CRFs/SAE Forms and the review of the data collection process. The FDA and regulatory authorities in other jurisdictions, including the IRB/IEC, may also request access to all study records, including source documentation, for inspection.

For sites participating in the study in the US, and in accordance with the Health Insurance Portability and Accountability Act (HIPAA) and associated regulations, an executed HIPAA authorization shall be obtained by the site from each subject (or the legal representative of the subject) before research activities may begin. Each HIPAA authorization shall comply with all HIPAA requirements including authorization allowing the site access to and use of the subject's personally identifiable health information, authorization for the site to disclose such information to Vertex, the FDA, and other parties requiring access under the protocol, and statements as to the purpose for which such information may be used and for how long.

#### 13.2.6 Record Retention

The investigator will maintain all study records according to ICH GCP guidelines and/or applicable local regulatory requirement(s), whichever is longest, as described in the Clinical Trial Agreement. If the investigator withdraws from the responsibility of keeping the study records, custody will be transferred to a person willing to accept the responsibility and Vertex will be notified.

## 13.2.7 Study Termination

At any time, Vertex may terminate this study in its entirety or may terminate this study at any particular site. In addition, for reasonable cause, either the investigators or their IRBs/IECs may terminate the study at their center.

Conditions that may lead to reasonable cause and warrant termination include, but are not limited to:

- Subject or investigator noncompliance
- Unsatisfactory subject enrollment
- Lack of adherence to protocol procedures
- Lack of evaluable and/or complete data
- Potentially unacceptable risk to study subjects
- Decision to modify drug development plan
- Decision by the FDA or other regulatory authority

Written notification that includes the reason for the clinical study termination is required.

#### 13.2.8 End of Study

The end of study is defined as the last scheduled visit or, for subjects who have been lost to follow-up, the last contact, whichever occurs later, for the latest completing subject in the study.

## 13.3 Data Quality Assurance

Vertex or its designated representative will conduct a study site visit to verify the qualifications of each investigator, inspect clinical study site facilities, and inform the investigator of responsibilities and procedures for ensuring adequate and correct study documentation.

The investigator is required to prepare and maintain adequate and accurate case histories designed to record all observations and other data pertinent to the study for each study participant. Study data for each enrolled subject will be entered into a CRF by study site personnel using a secure, validated, web-based electronic data capture (EDC) application. Vertex will have read-only access to site-entered clinical data in the EDC application.

Instances of missing, discrepant, or uninterpretable data will be queried with the investigator for resolution. Any changes to study data will be made to the CRF and documented in an audit trail, which will be maintained within the clinical database.

## 13.4 Monitoring

Monitoring and auditing procedures developed or approved by Vertex will be followed to comply with GCP guidelines. On-site checking of the CRFs/SAE Forms for completeness and clarity, cross-checking with source documents, and clarification of administrative matters will be performed.

The study will be monitored by Vertex or its designee. Monitoring will be done by personal visits from a representative of Vertex, or designee (study site monitor), who will review the CRFs/SAE Forms and source documents. The study site monitor will ensure that the investigation is conducted according to the protocol design and regulatory requirements.

Protocol deviations will be monitored and identified throughout study conduct as outlined in the Protocol Deviation Plan.

#### 13.5 Electronic Data Capture

Vertex will provide the study sites with secure access to and training on the EDC application sufficient to permit study site personnel to enter or correct information in the CRFs on the subjects for which they are responsible.

A CRF will be completed for each enrolled study subject. It is the investigator's responsibility to ensure the accuracy, completeness, clarity, and timeliness of the data reported in the subject's CRF. Source documentation supporting the CRF data will indicate the subject's participation in the study and will document the dates and details of study procedures, AEs, other observations, and subject status.

The investigator, or designated representative, will complete the CRF as soon as possible after information is collected.

The audit trail entry will show the user's identification information and the date and time of any correction. The investigator will provide formal approval of all the information in the CRFs, including any changes made to the CRFs, to endorse the final submitted data for the subjects for whom the investigator is responsible.

Vertex will retain the CRF data and corresponding audit trails. A copy of the final archival CRF in the form of a compact disc or other electronic media will be placed in the investigator's study file.

## 13.6 Publications and Clinical Study Report



## 13.6.2 Clinical Study Report

A CSR, written in accordance with the ICH E3 Guideline, will be submitted in accordance with local regulations.

#### 14 REFERENCES

- 1 Cystic Fibrosis Foundation. What is cystic fibrosis? Available at: https://www.cff.org/What-is-CF/About-Cystic-Fibrosis/. Accessed 03 September 2015.
- 2 Cystic Fibrosis Foundation. Patient Registry: 2014 Annual Data Report. Bethesda, MD: Cystic Fibrosis Foundation; 2015.
- European Cystic Fibrosis Society. 2013 ECFS Patient Registry Annual Data Report. Karup, Denmark: European Cystic Fibrosis Society; 2016.
- United States Department of Health and Human Services. Food and Drug Administration. Office of Orphan Products Development. Developing Products for Rare Diseases & Conditions. Available at: http://www.fda.gov/ForIndustry/DevelopingProductsforRareDiseasesConditions/default. htm. Accessed 19 September 2016.
- European Medicines Agency [Internet]. Committee for Orphan Medicinal Products (COMP). Available at:

  http://www.ema.europa.eu/ema/index.jsp?curl=pages/about\_us/general/general\_content\_
  000263.jsp&murl=menus/about\_us/about\_us.jsp&mid=WC0b01ac0580028e30.

  Accessed 19 September 2016.
- 6 Cystic Fibrosis Trust. UK Cystic Fibrosis Registry: Annual Data Report 2014. Bromley, Kent, UK: Cystic Fibrosis Trust; 2015.
- Flume PA, VanDevanter DR. State of progress in treating cystic fibrosis respiratory disease. BMC Med. 2012;10(1):88.
- 8 CFTR2.org. Clinical and functional translation of CFTR. The Clinical and Functional TRanslation of CFTR (CFTR2), US Cystic Fibrosis Foundation, Johns Hopkins University, the Hospital for Sick Children. Available at: http://www.cftr2.org. Accessed 19 July 2017.
- Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall GL, Culver BH, et al. Multi-ethnic reference values for spirometry for the 3–95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012;40(6):1324-43.
- Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, et al. Standardisation of spirometry. Eur Respir J. 2005;26(2):319-38.
- Levey AS, Bosch JP, Lewis JB, Greene T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation.

  Modification of Diet in Renal Disease Study Group. Ann Intern Med. 1999;130(6):461-70.
- Levey AS, Coresh J, Greene T, Stevens LA, Zhang YL, Hendriksen S, et al. Using standardized serum creatinine values in the modification of diet in renal disease study equation for estimating glomerular filtration rate. Ann Intern Med. 2006;145(4):247-54.
- 13 Counahan R, Chantler C, Ghazali S, Kirkwood B, Rose F, Barratt TM. Estimation of glomerular filtration rate from plasma creatinine concentration in children. Arch Dis Child. 1976;51(11):875-78.
- 14 Vertex Pharmaceuticals Incorporated. Tezacaftor (VX-661) Investigator's Brochure, Version 8 0 Report date: 07 November 2016

- Goss CH, Quittner AL. Patient-reported outcomes in cystic fibrosis. Proc Am Thorac
  - Goss CH, Quittner AL. Patient-reported outcomes in cystic fibrosis. Proc Am Thorac Soc. 2007;4(4):378-86.
  - 19 Quittner AL, Buu A, Messer MA, Modi AC, Watrous M. Development and validation of the Cystic Fibrosis Questionnaire in the United States. Chest. 2005;128(4):2347-54.
  - Henry B, Aussage P, Grosskopf C, Goehrs JM. Development of the Cystic Fibrosis Questionnaire (CFQ) for assessing quality of life in pediatric and adult patients. Qual Life Res. 2003;12(1):63-76.
  - Wenninger K, Aussage P, Wahn U, Staab D, German Cystic Fibrosis Questionnaire study group. The revised German Cystic Fibrosis Questionnaire: validation of a disease-specific health-related quality of life instrument. Qual Life Res. 2003;12(1):77-85.

## 15 PROTOCOL SIGNATURE PAGES

## 15.1 Sponsor Signature Page

| Protocol #: | VX17-659-103 | Version #: | 3.0 | Version Date: | 27 April 2018 |
|---|---|---|---|---|---|
| Study Title: A Phase 3, Randomized, Double-blind, Controlled Study Evaluating the Efficacy | | | | | |
| and Safety of VX-659 Combination Therapy in Subjects With Cystic Fibrosis Who Are | | | | | |
| Homozygous for the F508del Mutation (F/F) | | | | | |

This Clinical Study Protocol has been reviewed and approved by the sponsor.



## 15.2 Investigator Signature Page

| Protocol #: | VX17-659-103 | Version #: | 3.0 | Version Date: | 27 April 2018 |
|---|---|---|---|---|---|
| Study Title: A Phase 3, Randomized, Double-blind, Controlled Study Evaluating the Efficacy and Safety of VX-659 Combination Therapy in Subjects With Cystic Fibrosis Who Are Homozygous for the <i>F508del</i> Mutation (F/F) | | | | | |
| I have read Protocol VX17-659-103, Version 3.0, and agree to conduct the study according to its terms. I understand that all information concerning VX-659, tezacaftor, and ivacaftor and this protocol supplied to me by Vertex Pharmaceuticals Incorporated (Vertex) is confidential. | | | | | |
| Printed Name | | | _ | | |
| Signature | | | Date | 2 | |